CLINICAL TRIAL: NCT00153062
Title: PRoFESS - Prevention Regimen For Effectively Avoiding Second Strokes: A Double-blind, Active and Placebo Controlled Study of Aggrenox vs. Clopidogrel, With and Without Micardis
Brief Title: PRoFESS - Prevention Regimen For Effectively Avoiding Second Strokes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: GlaxoSmithKline (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9.159
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Aspirin, Dipyridamole Drug Combination; Telmisartan; Clopidogrel

ARMS (4):
- Aggrenox, Clopidogrel placebo, Micardis (Placebo Comparator): Aggrenox (25mg/200mg) bid, clopidogrel placebo qd, Micardis (80mg) qd
  Interventions: Drug: Aggrenox; Drug: Clopidogrel placebo; Drug: Micardis
- Aggrenox placebo, clopidogrel,, Micardis (Placebo Comparator): Clopidogrel (75mg) qd; Aggrenox placebo bid, Micardis (80mg) qd
  Interventions: Drug: Micardis; Drug: Aggrenox placebo; Drug: Clopidogrel
- Aggrenox, clop placebo, micardis placebo (Placebo Comparator): Aggrenox (25mg/200mg) bid, clopidogrel placebo qd, Micardis placebo qd
  Interventions: Drug: Aggrenox; Drug: Clopidogrel placebo; Drug: Micardis placebo
- Aggrenox plcebo, clop, micardis placebo (Placebo Comparator): Clopidogrel (75mg) qd, Aggrenox placebo bid, Micardis placebo qd.
  Interventions: Drug: Aggrenox placebo; Drug: Clopidogrel; Drug: Micardis placebo

INTERVENTIONS:
Drug: Aggrenox — 25mg aspirin, 200 mg dipyridamole
  Arms: Aggrenox, Clopidogrel placebo, Micardis
Drug: Aggrenox — 25mg aspirin, 200 mg dipyridamole
  Arms: Aggrenox, clop placebo, micardis placebo
Drug: Clopidogrel placebo — placebo
  Arms: Aggrenox, Clopidogrel placebo, Micardis
Drug: Clopidogrel placebo — placebo
  Arms: Aggrenox, clop placebo, micardis placebo
Drug: Micardis — 80 mg micardis
  Arms: Aggrenox, Clopidogrel placebo, Micardis
Drug: Micardis — 80 mg micardis
  Arms: Aggrenox placebo, clopidogrel,, Micardis
Drug: Aggrenox placebo — placebo
  Arms: Aggrenox placebo, clopidogrel,, Micardis
Drug: Aggrenox placebo — placebo
  Arms: Aggrenox plcebo, clop, micardis placebo
Drug: Clopidogrel — 75 mg clopidogrel
  Arms: Aggrenox placebo, clopidogrel,, Micardis
Drug: Clopidogrel — 75 mg clopidogrel
  Arms: Aggrenox plcebo, clop, micardis placebo
Drug: Micardis placebo — placebo
  Arms: Aggrenox, clop placebo, micardis placebo
Drug: Micardis placebo — placebo
  Arms: Aggrenox plcebo, clop, micardis placebo

SUMMARY:
The purpose of the trial is to determine if extended-release dipyridamole + aspirin [Aggrenox, Asasa ntin] is superior to clopidogrel [Plavix], and if telmisartan [Micardis, Gliosartan, Kinzal, Kinzalm ono, Predxal, Pritor, Samertan, Telmisartan] is superior to placebo, in the presence of background antihypertensive therapy, in prevention of a second stroke in patients who have recently suffered a stroke and therefore are at high risk of suffering another one.

ELIGIBILITY:
Inclusion criteria:

Male or female subjects 55 year or older who have suffered an ischemic stroke within the past 90 days and who meet all other inclusion criteria. Include also patients of ages 50 - 54 years and/or 90 to 120 days after the qualifying stroke provided the patient has at least two of the following additional risk factors:

* Diabetes mellitus
* Hypertension (systolic BP ¿ 140 or diastolic BP ¿ 90)
* Smoker at time of qualifying stroke
* Obesity (BMI>30; BMI=weight (kg)/[height (m)]2)
* Previous vascular disease (stroke, MI, or peripheral arterial disease prior to qualifying stroke)
* End-organ-damage (retinopathy, LVH, or microalbuminuria)
* Hyperlipidemia

Exclusion criteria:

hemorrhagic stroke (must be ruled out by imaging);unable to give informed consent; known brain tumor, severe renal or hepatic insufficiency, current active peptic ulcer disease, severe coronary artery disease including unstable angina pectoris or an MI within the previous 3 months,or history of a hemostatic disorder or systemic bleeding ;hyperkalemia;uncorrected volume or sodium depletion; pre-stroke history of dementia;modified Rankin score greater than 4;qualifying stroke induced by surgical or cardiovascular procedure;uncontrolled hypertension at entry above 180/110 mmHg (goal BPs are lower); SBP 120 mmHg or less for hospitalized patients; currently taking an ARB and not able or willing to switch to alternative; required or planned continuing treatment with antithrombotics or anticoagulants including heparin or warfarin or non-study platelet inhibitors; syndrome of asthma, rhinitis and nasal polyps;scheduled for major surgery, carotid endarterectomy, or carotid angioplasty (4 weeks post surgery is allowed);unlikely to be released from hospital following the qualifying stroke or presence of a severe disability likely to lead to being bedridden or demented or a non-vascular disease or condition which makes it unlikely that the patient will survive to the end of the trial; history of thrombocytopenia or neutropenia.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20332 (Actual)
Dates: Start 2003-08; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (667):
- United States (204):
  - 9.159.1101 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 9.159.1173 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 9.159.1058 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 9.159.1087 Boehringer Ingelheim Investigational Site, Montgomery, Alabama
  - 9.159.1081 Boehringer Ingelheim Investigational Site, Northport, Alabama
  - 9.159.1022 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 9.159.1133 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 9.159.1149 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 9.159.1137 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 9.159.1184 Boehringer Ingelheim Investigational Site, Fayetteville, Arkansas
  - 9.159.1005 Boehringer Ingelheim Investigational Site, Fort Smith, Arkansas
  - 9.159.1136 Boehringer Ingelheim Investigational Site, Jonesboro, Arkansas
  - 9.159.1062 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 9.159.1040 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 9.159.1180 Boehringer Ingelheim Investigational Site, Carmichael, California
  - 9.159.1114 Boehringer Ingelheim Investigational Site, Irvine, California
  - 9.159.1202 Boehringer Ingelheim Investigational Site, Laguna Hills, California
  - 9.159.1036 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 9.159.1052 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 9.159.1100 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 9.159.1111 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 9.159.1165 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 9.159.1134 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 9.159.1002 Boehringer Ingelheim Investigational Site, Palo Alto, California
  - 9.159.1108 Boehringer Ingelheim Investigational Site, Redding, California
  - 9.159.1013 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 9.159.1198 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 9.159.1029 Boehringer Ingelheim Investigational Site, San Diego, California
  - 9.159.1185 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 9.159.1218 Boehringer Ingelheim Investigational Site, San Jose, California
  - 9.159.1179 Boehringer Ingelheim Investigational Site, Santa Rosa, California
  - 9.159.1162 Boehringer Ingelheim Investigational Site, Sylmar, California
  - 9.159.1183 Boehringer Ingelheim Investigational Site, Torrance, California
  - 9.159.1205 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 9.159.1118 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 9.159.1045 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 9.159.1038 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 9.159.1196 Boehringer Ingelheim Investigational Site, Fairfield, Connecticut
  - 9.159.1018 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 9.159.1080 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 9.159.1120 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 9.159.1216 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 9.159.1057 Boehringer Ingelheim Investigational Site, Bay Pines, Florida
  - 9.159.1217 Boehringer Ingelheim Investigational Site, Boca Raton, Florida
  - 9.159.1096 Boehringer Ingelheim Investigational Site, Bradenton, Florida
  - 9.159.1144 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 9.159.1007 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 9.159.1190 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 9.159.1150 Boehringer Ingelheim Investigational Site, Ocala, Florida
  - 9.159.1153 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 9.159.1041 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 9.159.1072 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 9.159.1063 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 9.159.1208 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 9.159.1049 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 9.159.1176 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 9.159.1071 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 9.159.1079 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 9.159.1181 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 9.159.1138 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 9.159.1070 Boehringer Ingelheim Investigational Site, Rome, Georgia
  - 9.159.1107 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 9.159.1189 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 9.159.1026 University of Illinois, Chicago, Illinois
  - 9.159.1033 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 9.159.1060 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 9.159.1044 Boehringer Ingelheim Investigational Site, Maywood, Illinois
  - 9.159.1054 Boehringer Ingelheim Investigational Site, Palos Heights, Illinois
  - 9.159.1068 Boehringer Ingelheim Investigational Site, Park Ridge, Illinois
  - 9.159.1178 Boehringer Ingelheim Investigational Site, Peoria, Illinois
  - 9.159.1156 Boehringer Ingelheim Investigational Site, Elkhart, Indiana
  - 9.159.1092 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 9.159.1027 Boehringer Ingelheim Investigational Site, Cedar Rapids, Iowa
  - 9.159.1119 Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - 9.159.1187 Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - 9.159.1059 Boehringer Ingelheim Investigational Site, Iowa City, Iowa
  - 9.159.1135 Boehringer Ingelheim Investigational Site, Waterloo, Iowa
  - 9.159.1090 Boehringer Ingelheim Investigational Site, Kansas City, Kansas
  - 9.159.1129 Central Baptis Hospital, Lexington, Kentucky
  - 9.159.1131 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 9.159.1206 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 9.159.1212 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 9.159.1091 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 9.159.1147 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 9.159.1106 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 9.159.1194 Boehringer Ingelheim Investigational Site, Marrero, Louisiana
  - 9.159.1083 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 9.159.1195 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 9.159.1024 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 9.159.1055 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 9.159.1139 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 9.159.1031 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 9.159.1066 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 9.159.1104 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 9.159.1166 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 9.159.1192 Boehringer Ingelheim Investigational Site, South Weymouth, Massachusetts
  - 9.159.1039 Boehringer Ingelheim Investigational Site, Worchester, Massachusetts
  - 9.159.1019 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 9.159.1048 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 9.159.1089 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 9.159.1078 Boehringer Ingelheim Investigational Site, East Lansing, Michigan
  - 9.159.1143 Boehringer Ingelheim Investigational Site, Grand Rapids, Michigan
  - 9.159.1102 Boehringer Ingelheim Investigational Site, Kalamazoo, Michigan
  - 9.159.1011 Boehringer Ingelheim Investigational Site, Saginaw, Michigan
  - 9.159.1132 Boehringer Ingelheim Investigational Site, Southfield, Michigan
  - 9.159.1088 Boehringer Ingelheim Investigational Site, Duluth, Minnesota
  - 9.159.1158 Boehringer Ingelheim Investigational Site, Duluth, Minnesota
  - 9.159.1084 Boehringer Ingelheim Investigational Site, Golden Valley, Minnesota
  - 9.159.1097 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 9.159.1113 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 9.159.1128 St. Luke's Hospital MABSI Research, Kansas City, Missouri
  - 9.159.1172 Boehringer Ingelheim Investigational Site, Lees Summit, Missouri
  - 9.159.1009 Boehringer Ingelheim Investigational Site, Springfield, Missouri
  - 9.159.1174 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 9.159.1182 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 9.159.1191 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 9.159.1146 Boehringer Ingelheim Investigational Site, Great Falls, Montana
  - 9.159.1201 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 9.159.1127 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 9.159.1188 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 9.159.1204 Boehringer Ingelheim Investigational Site, Camden, New Jersey
  - 9.159.1203 Boehringer Ingelheim Investigational Site, Edison, New Jersey
  - 9.159.1042 Neurology Consultants of Burlington County, Lumberton, New Jersey
  - 9.159.1209 Boehringer Ingelheim Investigational Site, New Brunswick, New Jersey
  - 9.159.1125 Boehringer Ingelheim Investigational Site, Newark, New Jersey
  - 9.159.1095 Boehringer Ingelheim Investigational Site, Ridgewood, New Jersey
  - 9.159.1170 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 9.159.1086 Boehringer Ingelheim Investigational Site, Albany, New York
  - 9.159.1017 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 9.159.1064 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 9.159.1186 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 9.159.1151 Boehringer Ingelheim Investigational Site, Buffalo, New York
  - 9.159.1076 North Shore University Hospital, Manasset, New York
  - 9.159.1037 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 9.159.1220 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 9.159.1001 Boehringer Ingelheim Investigational Site, New York, New York
  - 9.159.1116 Boehringer Ingelheim Investigational Site, New York, New York
  - 9.159.1142 Saint Luke's-Roosevelt Hospital, New York, New York
  - 9.159.1126 Boehringer Ingelheim Investigational Site, Schenectady, New York
  - 9.159.1163 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 9.159.1121 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 9.159.1130 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 9.159.1169 Boehringer Ingelheim Investigational Site, Tonawanda, New York
  - 9.159.1065 Boehringer Ingelheim Investigational Site, White Plains, New York
  - 9.159.1099 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 9.159.1046 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 9.159.1094 Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - 9.159.1012 Boehringer Ingelheim Investigational Site, High Point, North Carolina
  - 9.159.1115, Wilmington, North Carolina
  - 9.159.1051 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 9.159.1110 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 9.159.1215 Boehringer Ingelheim Investigational Site, Bismarck, North Dakota
  - 9.159.1152 Boehringer Ingelheim Investigational Site, Fargo, North Dakota
  - 9.159.1159 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 9.159.1085 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 9.159.1032 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 9.159.1025 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 9.159.1177 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 9.159.1008 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 9.159.1141 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 9.159.1053 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 9.159.1122 Boehringer Ingelheim Investigational Site, Youngstown, Ohio
  - 9.159.1199 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 9.159.1010 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 9.159.1171 Boehringer Ingelheim Investigational Site, Abington, Pennsylvania
  - 9.159.1210 Boehringer Ingelheim Investigational Site, Allentown, Pennsylvania
  - 9.159.1214 Boehringer Ingelheim Investigational Site, Allentown, Pennsylvania
  - 9.159.1200 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 9.159.1043 Boehringer Ingelheim Investigational Site, Greensburg, Pennsylvania
  - 9.159.1164 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 9.159.1175 Boehringer Ingelheim Investigational Site, Lancaster, Pennsylvania
  - 9.159.1016 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 9.159.1056 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 9.159.1074 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 9.159.1112 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 9.159.1148 Boehringer Ingelheim Investigational Site, Upland, Pennsylvania
  - 9.159.1123 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 9.159.1140 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 9.159.1207 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 9.159.1004 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 9.159.1006 Boehringer Ingelheim Investigational Site, Bristol, Tennessee
  - 9.159.1154 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 9.159.1213 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 9.159.1075 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 9.159.1219 Boehringer Ingelheim Investigational Site, Brownwood, Texas
  - 9.159.1155 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 9.159.1197 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 9.159.1020 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 9.159.1023 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 9.159.1082 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 9.159.1160 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 9.159.1047 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 9.159.1069 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 9.159.1003 Boehringer Ingelheim Investigational Site, Bountiful, Utah
  - 9.159.1077 Boehringer Ingelheim Investigational Site, Newport News, Virginia
  - 9.159.1021 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 9.159.1061 Boehringer Ingelheim Investigational Site, Salem, Virginia
  - 9.159.1014 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 9.159.1145 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 9.159.1211 Boehringer Ingelheim Investigational Site, Charleston, West Virginia
  - 9.159.1035 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
  - 9.159.1030 Boehringer Ingelheim Investigational Site, Marshfield, Wisconsin
  - 9.159.1117 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
  - 9.159.1098 Community Healthcare Clinic Westhill Medical Specialists, Wausau, Wisconsin
- Argentina (7):
  - 9.159.1331 Boehringer Ingelheim Investigational Site, Capital Federal
  - 9.159.1333 Boehringer Ingelheim Investigational Site, Capital Federal
  - 9.159.1334 Boehringer Ingelheim Investigational Site, Capital Federal
  - 9.159.1335 Boehringer Ingelheim Investigational Site, Capital Federal
  - 9.159.1336 Boehringer Ingelheim Investigational Site, Capital Federal
  - 9.159.1332 Boehringer Ingelheim Investigational Site, Rosario, Santa Fe
  - 9.159.1342 Boehringer Ingelheim Investigational Site, Santa Fe
- Australia (10):
  - 9.159.2444 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 9.159.2449 Boehringer Ingelheim Investigational Site, New Lambton, New South Wales
  - 9.159.2448 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 9.159.2450 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 9.159.2452 Boehringer Ingelheim Investigational Site, Southport, Queensland
  - 9.159.2451 Boehringer Ingelheim Investigational Site, Bedford Park, South Australia
  - 9.159.2443 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 9.159.2447 Boehringer Ingelheim Investigational Site, Melbourne, Victoria
  - 9.159.2445 Boehringer Ingelheim Investigational Site, Parkville, Victoria
  - 9.159.2446 Boehringer Ingelheim Investigational Site, West Heidelberg, Victoria
- Austria (7):
  - 9.159.1515 Boehringer Ingelheim Investigational Site, Graz
  - 9.159.1519 Boehringer Ingelheim Investigational Site, Graz
  - 9.159.1517 Boehringer Ingelheim Investigational Site, Innsbruck
  - 9.159.1516 Boehringer Ingelheim Investigational Site, Linz
  - 9.159.1518 Boehringer Ingelheim Investigational Site, Ma.Gugging/Klosterneuburg
  - 9.159.1520 Boehringer Ingelheim Investigational Site, Sankt Pölten
  - 9.159.1521 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (14):
  - 9.159.1553 Boehringer Ingelheim Investigational Site, Aalst
  - 9.159.1543 Boehringer Ingelheim Investigational Site, Anderlecht
  - 9.159.1552 Boehringer Ingelheim Investigational Site, Antwerp
  - 9.159.1546 Boehringer Ingelheim Investigational Site, Bonheiden
  - 9.159.1547 Boehringer Ingelheim Investigational Site, Bruges
  - 9.159.1550 Boehringer Ingelheim Investigational Site, Brussels
  - 9.159.1549 Boehringer Ingelheim Investigational Site, Hasselt
  - 9.159.1555 Boehringer Ingelheim Investigational Site, Kortrijk
  - 9.159.1554 Boehringer Ingelheim Investigational Site, La Louvière
  - 9.159.1544 Boehringer Ingelheim Investigational Site, Leuven
  - 9.159.1548 Boehringer Ingelheim Investigational Site, Montegnée
  - 9.159.1556 Boehringer Ingelheim Investigational Site, Ottignies
  - 9.159.1545 Boehringer Ingelheim Investigational Site, Wilrijk
  - 9.159.1551 Boehringer Ingelheim Investigational Site, Yvoir
- Brazil (2):
  - 9.159.2869 Complexo Hospitalar Universitario Prof Edgard Santos, Salvador
  - 9.159.2853 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (42):
  - 9.159.1397 Foothills Medical Centre, Calgary, Alberta
  - 9.159.1382 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 9.159.1390 Boehringer Ingelheim Investigational Site, Lethbridge, Alberta
  - 9.159.1370 Boehringer Ingelheim Investigational Site, Kamloops, British Columbia
  - 9.159.1368 Boehringer Ingelheim Investigational Site, New Westminster, British Columbia
  - 9.159.1376 Boehringer Ingelheim Investigational Site, Penticton, British Columbia
  - 9.159.1387 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 9.159.1377 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 9.159.1355 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 9.159.1394 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 9.159.1356 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 9.159.1392 Boehringer Ingelheim Investigational Site, Corner Brook, Newfoundland and Labrador
  - 9.159.1385 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 9.159.1373 Boehringer Ingelheim Investigational Site, Sydney, Nova Scotia
  - 9.159.1393 Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - 9.159.1395 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 9.159.1360 Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - 9.159.1367 Boehringer Ingelheim Investigational Site, London, Ontario
  - 9.159.1384 Boehringer Ingelheim Investigational Site, London, Ontario
  - 9.159.1380 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 9.159.1378 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 9.159.1381 Ottawa Hospital General Campus, Ottawa, Ontario
  - 9.159.1366 Boehringer Ingelheim Investigational Site, Richmond Hill, Ontario
  - 9.159.1365 Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 9.159.1375 Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 9.159.1391 Boehringer Ingelheim Investigational Site, Tecumseh, Ontario
  - 9.159.1369 Boehringer Ingelheim Investigational Site, Thunder Bay, Ontario
  - 9.159.1357 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 9.159.1379 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 9.159.1383 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 9.159.1363 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 9.159.1359 Boehringer Ingelheim Investigational Site, Greenfield Park, Quebec
  - 9.159.1361 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 9.159.1362 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 9.159.1371 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 9.159.1374 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 9.159.1388 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 9.159.1372 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 9.159.1358 Boehringer Ingelheim Investigational Site, Saguenay, Quebec
  - 9.159.1364 Boehringer Ingelheim Investigational Site, Saint-Jérôme, Quebec
  - 9.159.1389 Boehringer Ingelheim Investigational Site, Regina, Saskatchewan
  - 9.159.1396 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (38):
  - 9.159.2490 Boehringer Ingelheim Investigational Site, Beijing
  - 9.159.2491 Boehringer Ingelheim Investigational Site, Beijing
  - 9.159.2492 Boehringer Ingelheim Investigational Site, Beijing
  - 9.159.2493 Boehringer Ingelheim Investigational Site, Beijing
  - 9.159.2494 Boehringer Ingelheim Investigational Site, Beijing
  - 9.159.2495 Boehringer Ingelheim Investigational Site, Beijing
  - 9.159.2496 Boehringer Ingelheim Investigational Site, Beijing
  - 9.159.2503 Boehringer Ingelheim Investigational Site, Changchun, Jilin Province
  - 9.159.2500 Boehringer Ingelheim Investigational Site, Changsha, Hunan Province
  - 9.159.2513 Boehringer Ingelheim Investigational Site, Chengdu, Sichuan Province
  - 9.159.2512 Boehringer Ingelheim Investigational Site, Chongqing
  - 9.159.2509 Boehringer Ingelheim Investigational Site, Guangzhou
  - 9.159.2518 Boehringer Ingelheim Investigational Site, Guangzhou
  - 9.159.2521 Boehringer Ingelheim Investigational Site, Guangzhou
  - 9.159.2507 Boehringer Ingelheim Investigational Site, Guangzhou, Guangdong Province
  - 9.159.2510 Boehringer Ingelheim Investigational Site, Guangzhou, Guangdong Province
  - 9.159.2502 Boehringer Ingelheim Investigational Site, Hangzhou, Zhejiang Province
  - 9.159.2504 Boehringer Ingelheim Investigational Site, Harbin, Heilongjiang Province
  - 9.159.2505 Boehringer Ingelheim Investigational Site, Jinan, Shandong Province
  - 9.159.2506 Boehringer Ingelheim Investigational Site, Jinan, Shangdong Province
  - 9.159.2517 Boehringer Ingelheim Investigational Site, Nanjing, Jiangsu Province
  - 9.159.2519 Boehringer Ingelheim Investigational Site, Nanjing, Jiangsu Province
  - 9.159.2520 Boehringer Ingelheim Investigational Site, Nanjing, Jiangsu Province
  - 9.159.2483 Boehringer Ingelheim Investigational Site, Shanghai
  - 9.159.2484 Boehringer Ingelheim Investigational Site, Shanghai
  - 9.159.2485 Boehringer Ingelheim Investigational Site, Shanghai
  - 9.159.2486 Boehringer Ingelheim Investigational Site, Shanghai
  - 9.159.2487 Boehringer Ingelheim Investigational Site, Shanghai
  - 9.159.2488 Boehringer Ingelheim Investigational Site, Shanghai
  - 9.159.2489 Boehringer Ingelheim Investigational Site, Shanghai
  - 9.159.2516 Boehringer Ingelheim Investigational Site, Suzhou, Jiangsu Province
  - 9.159.2497 Boehringer Ingelheim Investigational Site, Tianjin
  - 9.159.2501 Boehringer Ingelheim Investigational Site, Wenzhou, Zhejiang Province
  - 9.159.2498 Boehringer Ingelheim Investigational Site, Wuhan, Hubei Province
  - 9.159.2499 Boehringer Ingelheim Investigational Site, Wuhan, Hubei Province
  - 9.159.2511 Boehringer Ingelheim Investigational Site, Xi'an
  - 9.159.2515 Boehringer Ingelheim Investigational Site, Xian, Shanxi Province
  - 9.159.2514 Boehringer Ingelheim Investigational Site, Xian, Shanxi
- Denmark (10):
  - 9.159.1636 Boehringer Ingelheim Investigational Site, Aarhuc C
  - 9.159.1635 Boehringer Ingelheim Investigational Site, Aarhus C
  - 9.159.1639 Boehringer Ingelheim Investigational Site, Esbjerg
  - 9.159.1634 Boehringer Ingelheim Investigational Site, Frederiksberg
  - 9.159.1637 Boehringer Ingelheim Investigational Site, Glostrup Municipality
  - 9.159.1640 Boehringer Ingelheim Investigational Site, Hellerup
  - 9.159.1638 Boehringer Ingelheim Investigational Site, Hvidovre
  - 9.159.1633 Boehringer Ingelheim Investigational Site, København NV
  - 9.159.1631 Boehringer Ingelheim Investigational Site, København Ø
  - 9.159.1632 Boehringer Ingelheim Investigational Site, Odense
- 9.159.2181 Boehringer Ingelheim Investigational Site, Oviedo, El Salvador
- Finland (5):
  - 9.159.1655 Boehringer Ingelheim Investigational Site, Helsinki
  - 9.159.1658 Boehringer Ingelheim Investigational Site, Kuopio
  - 9.159.1659 Boehringer Ingelheim Investigational Site, Lappeenranta
  - 9.159.1656 Boehringer Ingelheim Investigational Site, Oulu
  - 9.159.1657 Boehringer Ingelheim Investigational Site, Seinäjoki
- France (7):
  - 9.159.1680 Boehringer Ingelheim Investigational Site, Lille
  - 9.159.1683 Boehringer Ingelheim Investigational Site, Limoges
  - 9.159.1681 Boehringer Ingelheim Investigational Site, Marseille
  - 9.159.1679 Boehringer Ingelheim Investigational Site, Nancy
  - 9.159.1685 Boehringer Ingelheim Investigational Site, Paris
  - 9.159.1682 Boehringer Ingelheim Investigational Site, Poitiers
  - 9.159.1684 Boehringer Ingelheim Investigational Site, Tours
- Germany (33):
  - 9.159.1713 Boehringer Ingelheim Investigational Site, Bad Neustadt/Saale
  - 9.159.1736 Boehringer Ingelheim Investigational Site, Berlin
  - 9.159.1732 Boehringer Ingelheim Investigational Site, Braunschweig
  - 9.159.1726 Boehringer Ingelheim Investigational Site, Cloppenburg
  - 9.159.1737 Boehringer Ingelheim Investigational Site, Cologne
  - 9.159.1723 Boehringer Ingelheim Investigational Site, Dresden
  - 9.159.1728 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 9.159.1707 Boehringer Ingelheim Investigational Site, Essen
  - 9.159.1738 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 9.159.1720 Boehringer Ingelheim Investigational Site, Giessen
  - 9.159.1722 Boehringer Ingelheim Investigational Site, Hamburg
  - 9.159.1739 Boehringer Ingelheim Investigational Site, Hamburg
  - 9.159.1724 Boehringer Ingelheim Investigational Site, Heidelberg
  - 9.159.1734 Boehringer Ingelheim Investigational Site, Jena
  - 9.159.1730 Boehringer Ingelheim Investigational Site, Kaiserslautern
  - 9.159.1717 Boehringer Ingelheim Investigational Site, Leipzig
  - 9.159.1735 Boehringer Ingelheim Investigational Site, Ludwigshafen am Rhein
  - 9.159.1712 Boehringer Ingelheim Investigational Site, Magdeburg
  - 9.159.1710 Boehringer Ingelheim Investigational Site, Mainz
  - 9.159.1709 Boehringer Ingelheim Investigational Site, Minden
  - 9.159.1716 Boehringer Ingelheim Investigational Site, Mönchengladbach
  - 9.159.1718 Boehringer Ingelheim Investigational Site, München
  - 9.159.1725 Boehringer Ingelheim Investigational Site, München
  - 9.159.1729 Boehringer Ingelheim Investigational Site, München
  - 9.159.1727 Boehringer Ingelheim Investigational Site, Münster
  - 9.159.1711 Boehringer Ingelheim Investigational Site, Nuremberg
  - 9.159.1719 Boehringer Ingelheim Investigational Site, Regensburg
  - 9.159.1731 Boehringer Ingelheim Investigational Site, Remscheid
  - 9.159.1708 Boehringer Ingelheim Investigational Site, Rostock
  - 9.159.1715 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 9.159.1714 Boehringer Ingelheim Investigational Site, Siegen
  - 9.159.1733 Boehringer Ingelheim Investigational Site, Stuttgart
  - 9.159.1721 Boehringer Ingelheim Investigational Site, Weimar
- Greece (6):
  - 9.159.1826 Boehringer Ingelheim Investigational Site, Alexandroupoli
  - 9.159.1819 Boehringer Ingelheim Investigational Site, Athens
  - 9.159.1820 Boehringer Ingelheim Investigational Site, Athens
  - 9.159.1821 Boehringer Ingelheim Investigational Site, Athens
  - 9.159.1825 Boehringer Ingelheim Investigational Site, Ioannina
  - 9.159.1824 Boehringer Ingelheim Investigational Site, Pátrai
- Hong Kong (2):
  - 9.159.2713 Boehringer Ingelheim Investigational Site, Hong Kong
  - 9.159.2714 Boehringer Ingelheim Investigational Site, Hong Kong
- India (30):
  - 9.159.2605 Boehringer Ingelheim Investigational Site, Annāmalainagar
  - 9.159.2603 Boehringer Ingelheim Investigational Site, Bangalore
  - 9.159.2620 Boehringer Ingelheim Investigational Site, Bangalore
  - 9.159.2616 Boehringer Ingelheim Investigational Site, Bikaner
  - 9.159.2618 Boehringer Ingelheim Investigational Site, Calicut
  - 9.159.2604 Boehringer Ingelheim Investigational Site, Chennai
  - 9.159.2619 Boehringer Ingelheim Investigational Site, Chennai
  - 9.159.2625 Boehringer Ingelheim Investigational Site, Chennai
  - 9.159.2607 Boehringer Ingelheim Investigational Site, Hyderabad
  - 9.159.2624 Boehringer Ingelheim Investigational Site, Hyderabad
  - 9.159.2630 Boehringer Ingelheim Investigational Site, Hyderabad
  - 9.159.2632 Boehringer Ingelheim Investigational Site, Hyderabad
  - 9.159.2610 Boehringer Ingelheim Investigational Site, Indore
  - 9.159.2615 Boehringer Ingelheim Investigational Site, Jaipur
  - 9.159.2617 Boehringer Ingelheim Investigational Site, Jaipur
  - 9.159.2612 Boehringer Ingelheim Investigational Site, Jodhpur
  - 9.159.2606 Boehringer Ingelheim Investigational Site, Kochi
  - 9.159.2621 Boehringer Ingelheim Investigational Site, Kottayam
  - 9.159.2613 Boehringer Ingelheim Investigational Site, Lucknow
  - 9.159.2614 Boehringer Ingelheim Investigational Site, Ludhiana
  - 9.159.2611 Boehringer Ingelheim Investigational Site, Mumbai
  - 9.159.2628 Boehringer Ingelheim Investigational Site, New Delhi
  - 9.159.2629 Boehringer Ingelheim Investigational Site, New Delhi
  - 9.159.2623 Boehringer Ingelheim Investigational Site, Patiāla
  - 9.159.2609 Boehringer Ingelheim Investigational Site, Pune
  - 9.159.2622 Boehringer Ingelheim Investigational Site, Pune
  - 9.159.2627 Boehringer Ingelheim Investigational Site, Secunderabad
  - 9.159.2626 Boehringer Ingelheim Investigational Site, Trichy
  - 9.159.2631 Boehringer Ingelheim Investigational Site, Visakhapatnam
  - 9.159.2608 Boehringer Ingelheim Investigational Site, Wardha
- Ireland (2):
  - 9.159.1851 Boehringer Ingelheim Investigational Site, Cork
  - 9.159.1852 Boehringer Ingelheim Investigational Site, Dublin
- Israel (8):
  - 9.159.2729 Barzilai Medical Center, Ashkelon
  - 9.159.2721 Neurology Unit, Haifa
  - 9.159.2724 Rambam Medical Center, Tel-Aviv Medical, Haifa
  - 9.159.2723 Boehringer Ingelheim Investigational Site, Israel
  - 9.159.2727 Western Galilee Hospital, Nahariya
  - 9.159.2722 Neurology Unit, Petah Tikva
  - 9.159.2725 Tel Aviv Medical Center, Tel Aviv
  - 9.159.2726 Sheba Medical Center, Tel Litwinsky
- Italy (22):
  - 9.159.1875 Università degli Studi di Ancona, Ancona
  - 9.159.1882 Ospedale Brotzu, Cagliari
  - 9.159.1883 Azienda Ospedaliera S. Anna, Como
  - 9.159.1871 Azienda Ospedaliera "Careggi", Florence
  - 9.159.1869 Università degli Studi di Genova, Genova
  - 9.159.1870 ASL No. 5 di Jesi, Jesi (ancona)
  - 9.159.1865 Ospedale Regionale "S. Salvatore", L’Aquila
  - 9.159.1866 Ospedale S. Raffaele, Milan
  - 9.159.1873 Istituto Scientifico "S. Luca", Milan
  - 9.159.1884 Ospedale S. Carlo Borromeo", Milan
  - 9.159.1868 Ospedale "S. Maria di Loreto Mare", Napoli
  - 9.159.1876 Azienda Ospedaliera di Padova -Policlinico Universitario, Padua
  - 9.159.1874 Ospedale Civico - ARNAS, Palermo
  - 9.159.1872 Neuromed IRCCS, Pozzilli (IS)
  - 9.159.1879 Policlinico S. Andrea, Roma
  - 9.159.1881 Università "La Sapienza", Roma
  - 9.159.1877 Azienda Ospedaliera Umberto I, Syracuse
  - 9.159.1878 Azienda Ospedaliera "Santo Maria", Terni
  - 9.159.1864 Azienda Ospedaliera "S. Giovanni Battista", Torino
  - 9.159.1863 Ospedale di Cattinara, Trieste
  - 9.159.1867 Presidio Ospedaliero G.Jazzolino, Vibo Valentia
  - 9.159.1880 Ospedale Civile, Vicenza
- Japan (40):
  - 9.159.2964 Boehringer Ingelheim Investigational Site, Adachi-ku, Tokyo
  - 9.159.2958 Boehringer Ingelheim Investigational Site, Akashi, Hyogo
  - 9.159.2970 Boehringer Ingelheim Investigational Site, Akashi, Hyogo
  - 9.159.2965 Boehringer Ingelheim Investigational Site, Ako, Hyogo
  - 9.159.2968 Boehringer Ingelheim Investigational Site, Aoba-ku, Yokohama, Kanagawa
  - 9.159.2951 Boehringer Ingelheim Investigational Site, Azumino, Nagano
  - 9.159.2959 Boehringer Ingelheim Investigational Site, Chitose, Hokkaido
  - 9.159.2944 Boehringer Ingelheim Investigational Site, Chuo-ku, Kobe, Hyogo
  - 9.159.2947 Boehringer Ingelheim Investigational Site, Chuo-Ku, Sapporo, Hokkaido
  - 9.159.2954 Boehringer Ingelheim Investigational Site, Fushimi-ku, Kyoto, Kyoto
  - 9.159.2942 Boehringer Ingelheim Investigational Site, Habikino, Osaka
  - 9.159.2948 Boehringer Ingelheim Investigational Site, Higashi-ku, Sapporo, Hokkaido
  - 9.159.2957 Boehringer Ingelheim Investigational Site, Higashi-osaka, Osaka
  - 9.159.2940 Boehringer Ingelheim Investigational Site, Higashinari-ku, Osaka, Osaka
  - 9.159.2973 Boehringer Ingelheim Investigational Site, Higashiyodogawa-ku, Osaka, Osaka
  - 9.159.2949 Boehringer Ingelheim Investigational Site, Hitachinaka, Ibaraki
  - 9.159.2953 Boehringer Ingelheim Investigational Site, Iida, Nagano
  - 9.159.2943 Boehringer Ingelheim Investigational Site, Izumisano, Osaka
  - 9.159.2963 Boehringer Ingelheim Investigational Site, Jyonan-ku, Fukuoka, Fukuoka
  - 9.159.2933 Boehringer Ingelheim Investigational Site, Kasama, Ibaraki
  - 9.159.2955 Boehringer Ingelheim Investigational Site, Kasuga, Fukuoka
  - 9.159.2938 Boehringer Ingelheim Investigational Site, Kita-ku, Osaka, Osaka
  - 9.159.2967 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 9.159.2969 Boehringer Ingelheim Investigational Site, Kushiro
  - 9.159.2952 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 9.159.2961 Boehringer Ingelheim Investigational Site, Midori-ku, Yokohama, Kanagawa
  - 9.159.2934 Boehringer Ingelheim Investigational Site, Moriya, Ibaraki
  - 9.159.2971 Boehringer Ingelheim Investigational Site, Musashino, Tokyo
  - 9.159.2962 Boehringer Ingelheim Investigational Site, Nakagawa-ku, Nagoya, Aichi
  - 9.159.2939 Boehringer Ingelheim Investigational Site, Nishi-yodogawa-ku, Osaka, Osaka
  - 9.159.2956 Boehringer Ingelheim Investigational Site, Ohnojo, Fukuoka
  - 9.159.2941 Boehringer Ingelheim Investigational Site, Sakai-ku, Sakai, Osaka
  - 9.159.2945 Boehringer Ingelheim Investigational Site, Sawara-ku, Fukuoka, Fukuoka
  - 9.159.2937 Boehringer Ingelheim Investigational Site, Shimogyo-ku, Kyoto, Kyoto
  - 9.159.2966 Boehringer Ingelheim Investigational Site, Shiroishi, Miyagi
  - 9.159.2936 Boehringer Ingelheim Investigational Site, Suwa, Nagano
  - 9.159.2946 Boehringer Ingelheim Investigational Site, Takikawa, Hokkaido
  - 9.159.2935 Boehringer Ingelheim Investigational Site, Tatebayashi, Gunma
  - 9.159.2950 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaraki
  - 9.159.2972 Boehringer Ingelheim Investigational Site, Yao, Osaka
- Malaysia (2):
  - 9.159.2707 Boehringer Ingelheim Investigational Site, Kelantan Darul Naim
  - 9.159.2706 Boehringer Ingelheim Investigational Site, Kuala Lumpur
- 9.159.2765 Boehringer Ingelheim Investigational Site, Metepec, Mexico
- Netherlands (22):
  - 9.159.1960 Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - 9.159.1945 Medisch Centrum Alkmaar, Alkmaar
  - 9.159.1963 Polikliniek Neurologie, Assen
  - 9.159.1949 Ziekenhuis Gooi-Noord, Blaricum
  - 9.159.1962 Locatie Molengracht, Breda
  - 9.159.1959 Catharina Ziekenhuis, Eindhoven
  - 9.159.1946 Scheper Ziekenhuis, Emmen
  - 9.159.1958 Medisch Spectrum Twente, Enschede
  - 9.159.1943 Umcg, Groningen
  - 9.159.1961 Lokatie Van Swieten, Groningen
  - 9.159.1953 Atrium Medisch Centrum, Heerlen
  - 9.159.1955 Elkerliek Ziekenhuis, Helmond
  - 9.159.1951 Ziekenhuisgroep Twente, Hengelo
  - 9.159.1948 Medisch Centrum Leeuwarden, Leeuwarden
  - 9.159.1952 Rijnland Ziekenhuis, Leiderdorp
  - 9.159.1947 Sint Antonius Ziekenhuis, Nieuwegein
  - 9.159.1964 Canisius-Wilhelmina ziekenhuis, Nijmegen
  - 9.159.1950 HagaZiekenhuis, The Hague
  - 9.159.1956 TweeSteden Ziekenhuis Tilburg, Tilburg
  - 9.159.1957 Sint Elisabeth Ziekenhuis, Tilburg
  - 9.159.1944 Máxima Medisch Centrum, Veldhoven
  - 9.159.1954 St. Jans Gasthuis, Weert
- Norway (3):
  - 9.159.2029 Boehringer Ingelheim Investigational Site, Bergen
  - 9.159.2028 Boehringer Ingelheim Investigational Site, Oslo
  - 9.159.2027 Boehringer Ingelheim Investigational Site, Trondheim
- Portugal (4):
  - 9.159.2040 Hospital Fernando Fonseca, Amadora
  - 9.159.2039 Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - 9.159.2041 Centro Hospitalar de Lisboa Norte, Lisbon
  - 9.159.2042 Centro Hospitalar do Porto, Porto
- Russia (41):
  - 9.159.2102 Boehringer Ingelheim Investigational Site, Kazan'
  - 9.159.2117 Boehringer Ingelheim Investigational Site, Kemerovo
  - 9.159.2107 Boehringer Ingelheim Investigational Site, Kirov
  - 9.159.2116 Boehringer Ingelheim Investigational Site, Krasnoyarsk
  - 9.159.2079 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2080 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2081 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2082 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2083 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2084 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2085 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2087 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2088 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2089 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2090 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2091 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2092 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2093 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2095 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2098 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2101 Boehringer Ingelheim Investigational Site, Moscow
  - 9.159.2105 Boehringer Ingelheim Investigational Site, Nizhnyi Novgorod
  - 9.159.2115 Boehringer Ingelheim Investigational Site, Novosibirsk
  - 9.159.2119 Boehringer Ingelheim Investigational Site, Omsk
  - 9.159.2111 Boehringer Ingelheim Investigational Site, Oryol
  - 9.159.2106 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 9.159.2094 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 9.159.2097 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 9.159.2099 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 9.159.2100 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 9.159.2108 Boehringer Ingelheim Investigational Site, Samara
  - 9.159.2109 Boehringer Ingelheim Investigational Site, Saratov
  - 9.159.2110 Boehringer Ingelheim Investigational Site, Saratov
  - 9.159.2118 Boehringer Ingelheim Investigational Site, Seversk
  - 9.159.2086 Boehringer Ingelheim Investigational Site, Smolensk
  - 9.159.2120 Boehringer Ingelheim Investigational Site, Ufa
  - 9.159.2112 Boehringer Ingelheim Investigational Site, Volgograd
  - 9.159.2113 Boehringer Ingelheim Investigational Site, Volgograd
  - 9.159.2104 Boehringer Ingelheim Investigational Site, Voronezh
  - 9.159.2103 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 9.159.2114 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Singapore (3):
  - 9.159.2703 Boehringer Ingelheim Investigational Site, Singapore
  - 9.159.2704 Boehringer Ingelheim Investigational Site, Singapore
  - 9.159.2705 Boehringer Ingelheim Investigational Site, Singapore
- South Africa (7):
  - 9.159.2060 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 9.159.2056 Boehringer Ingelheim Investigational Site, Cape Town
  - 9.159.2057 Boehringer Ingelheim Investigational Site, Durban
  - 9.159.2055 Boehringer Ingelheim Investigational Site, Johannesburg
  - 9.159.2061 Boehringer Ingelheim Investigational Site, Johannesburg
  - 9.159.2058 Boehringer Ingelheim Investigational Site, Pretoria
  - 9.159.2059 Boehringer Ingelheim Investigational Site, Sunninghill
- South Korea (7):
  - 9.159.1593 Boehringer Ingelheim Investigational Site, Gwangju
  - 9.159.1595 Boehringer Ingelheim Investigational Site, Incheon
  - 9.159.1592 Boehringer Ingelheim Investigational Site, Kyunggi-do
  - 9.159.1591 Boehringer Ingelheim Investigational Site, Seoul
  - 9.159.1594 Boehringer Ingelheim Investigational Site, Seoul
  - 9.159.1597 Boehringer Ingelheim Investigational Site, Seoul
  - 9.159.1596 Boehringer Ingelheim Investigational Site, Suwon
- Spain (6):
  - 9.159.2179 Boehringer Ingelheim Investigational Site, Alicante
  - 9.159.2177 Boehringer Ingelheim Investigational Site, Barcelona
  - 9.159.2178 Boehringer Ingelheim Investigational Site, Hospitalet de Llobregat (Barcelona)
  - 9.159.2175 Boehringer Ingelheim Investigational Site, Madrid
  - 9.159.2176 Boehringer Ingelheim Investigational Site, Madrid
  - 9.159.2180 Boehringer Ingelheim Investigational Site, Pamplona
- Sweden (19):
  - 9.159.2223 Boehringer Ingelheim Investigational Site, Borås
  - 9.159.2209 Boehringer Ingelheim Investigational Site, Eskilstuna
  - 9.159.2204 Boehringer Ingelheim Investigational Site, Gothenburg
  - 9.159.2205 Boehringer Ingelheim Investigational Site, Gothenburg
  - 9.159.2728 Neurology Unit, Holon
  - 9.159.2210 Boehringer Ingelheim Investigational Site, Jönköping
  - 9.159.2206 Boehringer Ingelheim Investigational Site, Lund
  - 9.159.2211 Boehringer Ingelheim Investigational Site, Mora
  - 9.159.2208 Boehringer Ingelheim Investigational Site, Örebro
  - 9.159.2216 Boehringer Ingelheim Investigational Site, Skellefteå
  - 9.159.2215 Boehringer Ingelheim Investigational Site, Skövde
  - 9.159.2203 Boehringer Ingelheim Investigational Site, Stockholm
  - 9.159.2212 Boehringer Ingelheim Investigational Site, Stockholm
  - 9.159.2213 Boehringer Ingelheim Investigational Site, Stockholm
  - 9.159.2222 Boehringer Ingelheim Investigational Site, Stockholm
  - 9.159.2225 Boehringer Ingelheim Investigational Site, Stockholm
  - 9.159.2207 Boehringer Ingelheim Investigational Site, Umeå
  - 9.159.2214 Boehringer Ingelheim Investigational Site, Värnamo
  - 9.159.2224 Boehringer Ingelheim Investigational Site, Västervik
- Taiwan (12):
  - 9.159.2250 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 9.159.2253 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 9.159.2248 Boehringer Ingelheim Investigational Site, Taichung
  - 9.159.2249 Boehringer Ingelheim Investigational Site, Taichung
  - 9.159.2251 Boehringer Ingelheim Investigational Site, Tainan
  - 9.159.2244 Boehringer Ingelheim Investigational Site, Taipei
  - 9.159.2245 Boehringer Ingelheim Investigational Site, Taipei
  - 9.159.2246 Boehringer Ingelheim Investigational Site, Taipei
  - 9.159.2247 Boehringer Ingelheim Investigational Site, Taipei
  - 9.159.2252 Boehringer Ingelheim Investigational Site, Taipei
  - 9.159.2254 Boehringer Ingelheim Investigational Site, Taipei
  - 9.159.2243 Boehringer Ingelheim Investigational Site, Taoyuan District
- Thailand (5):
  - 9.159.2797 Boehringer Ingelheim Investigational Site, Bangkok
  - 9.159.2798 Boehringer Ingelheim Investigational Site, Bangkok
  - 9.159.2799 Boehringer Ingelheim Investigational Site, Bangkok
  - 9.159.2800 Boehringer Ingelheim Investigational Site, Bangkok
  - 9.159.2801 Boehringer Ingelheim Investigational Site, Chiang Mai
- Turkey (Türkiye) (7):
  - 9.159.2830 Boehringer Ingelheim Investigational Site, Ankara
  - 9.159.2829 Boehringer Ingelheim Investigational Site, Antalya
  - 9.159.2831 Boehringer Ingelheim Investigational Site, Bursa
  - 9.159.2827 Boehringer Ingelheim Investigational Site, Eskişehir
  - 9.159.2825 Boehringer Ingelheim Investigational Site, Istanbul
  - 9.159.2826 Boehringer Ingelheim Investigational Site, Istanbul
  - 9.159.2828 Dkuz Eylul Universitesi Tip Fakultesi Noroloji A.B.D., Izmir
- Ukraine (12):
  - 9.159.2387 Boehringer Ingelheim Investigational Site, Dnipro
  - 9.159.2384 Boehringer Ingelheim Investigational Site, Kharkiv
  - 9.159.2385 Boehringer Ingelheim Investigational Site, Kharkiv
  - 9.159.2386 Boehringer Ingelheim Investigational Site, Kharkiv
  - 9.159.2392 Boehringer Ingelheim Investigational Site, Kharkiv
  - 9.159.2379 Boehringer Ingelheim Investigational Site, Kyiv
  - 9.159.2380 Boehringer Ingelheim Investigational Site, Kyiv
  - 9.159.2382 Boehringer Ingelheim Investigational Site, Kyiv
  - 9.159.2389 Boehringer Ingelheim Investigational Site, Odesa
  - 9.159.2390 Boehringer Ingelheim Investigational Site, Odesa
  - 9.159.2391 Boehringer Ingelheim Investigational Site, Vinnytzya
  - 9.159.2388 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (26):
  - 9.159.2304 Boehringer Ingelheim Investigational Site, Belfast
  - 9.159.2297 Boehringer Ingelheim Investigational Site, Birmingham
  - 9.159.2299 Boehringer Ingelheim Investigational Site, Bournemouth
  - 9.159.2301 Boehringer Ingelheim Investigational Site, Bristol
  - 9.159.2298 Boehringer Ingelheim Investigational Site, Dundee
  - 9.159.2307 Boehringer Ingelheim Investigational Site, Exeter
  - 9.159.2296 Boehringer Ingelheim Investigational Site, Glasgow
  - 9.159.2300 Boehringer Ingelheim Investigational Site, Glasgow
  - 9.159.2287 Boehringer Ingelheim Investigational Site, Harrow
  - 9.159.2303 Boehringer Ingelheim Investigational Site, Henshingham, Whitehaven
  - 9.159.2308 Boehringer Ingelheim Investigational Site, Leicester
  - 9.159.2295 Boehringer Ingelheim Investigational Site, Liverpool
  - 9.159.2286 Boehringer Ingelheim Investigational Site, London
  - 9.159.2293 Boehringer Ingelheim Investigational Site, London
  - 9.159.2294 Boehringer Ingelheim Investigational Site, London
  - 9.159.2305 Boehringer Ingelheim Investigational Site, Mansfield
  - 9.159.2290 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 9.159.2288 Boehringer Ingelheim Investigational Site, North Shields
  - 9.159.2285 Boehringer Ingelheim Investigational Site, Northampton
  - 9.159.2284 Boehringer Ingelheim Investigational Site, Nottingham
  - 9.159.2283 Boehringer Ingelheim Investigational Site, Poole
  - 9.159.2302 Boehringer Ingelheim Investigational Site, Rotherham
  - 9.159.2292 Boehringer Ingelheim Investigational Site, Sheffield
  - 9.159.2289 Boehringer Ingelheim Investigational Site, Southampton
  - 9.159.2306 Boehringer Ingelheim Investigational Site, Stoke-on-Trent
  - 9.159.2291 Boehringer Ingelheim Investigational Site, Sunderland

REFERENCES:
- [Derived] Ovbiagele B, Bath PM, Cotton D, Sha N, Diener HC; PRoFESS Investigators. Low glomerular filtration rate, recurrent stroke risk, and effect of renin-angiotensin system modulation. Stroke. 2013 Nov;44(11):3223-5. doi: 10.1161/STROKEAHA.113.002463. Epub 2013 Aug 29. PMID 23988639
- [Derived] Bohm M, Cotton D, Foster L, Custodis F, Laufs U, Sacco R, Bath PM, Yusuf S, Diener HC. Impact of resting heart rate on mortality, disability and cognitive decline in patients after ischaemic stroke. Eur Heart J. 2012 Nov;33(22):2804-12. doi: 10.1093/eurheartj/ehs250. Epub 2012 Aug 26. PMID 22922507
- [Derived] Weber R, Weimar C, Blatchford J, Hermansson K, Wanke I, Moller-Hartmann C, Gizewski ER, Forsting M, Demchuk AM, Sacco RL, Saver JL, Warach S, Diener HC, Diehl A; PRoFESS Imaging Substudy Group. Telmisartan on top of antihypertensive treatment does not prevent progression of cerebral white matter lesions in the prevention regimen for effectively avoiding second strokes (PRoFESS) MRI substudy. Stroke. 2012 Sep;43(9):2336-42. doi: 10.1161/STROKEAHA.111.648576. Epub 2012 Jun 26. PMID 22738922
- [Derived] Weber R, Weimar C, Wanke I, Moller-Hartmann C, Gizewski ER, Blatchford J, Hermansson K, Demchuk AM, Forsting M, Sacco RL, Saver JL, Warach S, Diener HC, Diehl A; PRoFESS Imaging Substudy Group. Risk of recurrent stroke in patients with silent brain infarction in the Prevention Regimen for Effectively Avoiding Second Strokes (PRoFESS) imaging substudy. Stroke. 2012 Feb;43(2):350-5. doi: 10.1161/STROKEAHA.111.631739. Epub 2012 Jan 19. PMID 22267825
- [Derived] Ovbiagele B, Diener HC, Yusuf S, Martin RH, Cotton D, Vinisko R, Donnan GA, Bath PM; PROFESS Investigators. Level of systolic blood pressure within the normal range and risk of recurrent stroke. JAMA. 2011 Nov 16;306(19):2137-44. doi: 10.1001/jama.2011.1650. PMID 22089721
- [Derived] Diener HC, Sacco RL, Yusuf S, Cotton D, Ounpuu S, Lawton WA, Palesch Y, Martin RH, Albers GW, Bath P, Bornstein N, Chan BP, Chen ST, Cunha L, Dahlof B, De Keyser J, Donnan GA, Estol C, Gorelick P, Gu V, Hermansson K, Hilbrich L, Kaste M, Lu C, Machnig T, Pais P, Roberts R, Skvortsova V, Teal P, Toni D, VanderMaelen C, Voigt T, Weber M, Yoon BW; Prevention Regimen for Effectively Avoiding Second Strokes (PRoFESS) study group. Effects of aspirin plus extended-release dipyridamole versus clopidogrel and telmisartan on disability and cognitive function after recurrent stroke in patients with ischaemic stroke in the Prevention Regimen for Effectively Avoiding Second Strokes (PRoFESS) trial: a double-blind, active and placebo-controlled study. Lancet Neurol. 2008 Oct;7(10):875-84. doi: 10.1016/S1474-4422(08)70198-4. Epub 2008 Aug 29. PMID 18757238
- [Derived] Yusuf S, Diener HC, Sacco RL, Cotton D, Ounpuu S, Lawton WA, Palesch Y, Martin RH, Albers GW, Bath P, Bornstein N, Chan BP, Chen ST, Cunha L, Dahlof B, De Keyser J, Donnan GA, Estol C, Gorelick P, Gu V, Hermansson K, Hilbrich L, Kaste M, Lu C, Machnig T, Pais P, Roberts R, Skvortsova V, Teal P, Toni D, VanderMaelen C, Voigt T, Weber M, Yoon BW; PRoFESS Study Group. Telmisartan to prevent recurrent stroke and cardiovascular events. N Engl J Med. 2008 Sep 18;359(12):1225-37. doi: 10.1056/NEJMoa0804593. Epub 2008 Aug 27. PMID 18753639
- [Derived] Sacco RL, Diener HC, Yusuf S, Cotton D, Ounpuu S, Lawton WA, Palesch Y, Martin RH, Albers GW, Bath P, Bornstein N, Chan BP, Chen ST, Cunha L, Dahlof B, De Keyser J, Donnan GA, Estol C, Gorelick P, Gu V, Hermansson K, Hilbrich L, Kaste M, Lu C, Machnig T, Pais P, Roberts R, Skvortsova V, Teal P, Toni D, Vandermaelen C, Voigt T, Weber M, Yoon BW; PRoFESS Study Group. Aspirin and extended-release dipyridamole versus clopidogrel for recurrent stroke. N Engl J Med. 2008 Sep 18;359(12):1238-51. doi: 10.1056/NEJMoa0805002. Epub 2008 Aug 27. PMID 18753638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sept 2003 - July 2006; 695 centres in 35 countries
Pre-assignment Details: No screening period
Groups:
- Aspirin + Extended Release Dipyridamole / Telmisartan: 25 milligrams (mg) aspirin + 200 mg extended-release dipyridamole, twice daily, capsule / telmisartan 80 mg, once daily, tablet
- Aspirin + Extended Release Dipyridamole / Placebo: 25 mg aspirin + 200 mg extended-release dipyridamole, twice daily, capsule / placebo tablet
- Clopidogrel / Telmisartan: clopidogrel 75 mg, once daily, tablet / telmisartan 80 mg, once daily, tablet
- Clopidogrel / Placebo: clopidogrel 75 mg, once daily, tablet / placebo tablet
Period: Overall Study
Arm/Group | Aspirin + Extended Release Dipyridamole / Telmisartan | Aspirin + Extended Release Dipyridamole / Placebo | Clopidogrel / Telmisartan | Clopidogrel / Placebo
Started | 5086 | 5095 | 5060 | 5091
Completed | 4699 | 4689 | 4645 | 4680
Not Completed | 387 | 406 | 415 | 411
Not completed — Death | 360 | 352 | 369 | 365
Not completed — Withdrawal by Subject | 14 | 30 | 27 | 28
Not completed — Lost to Follow-up | 12 | 20 | 15 | 16
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 1 | 1
Not completed — No disposition data available | 1 | 1 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin + Extended Release Dipyridamole / Telmisartan | Aspirin + Extended Release Dipyridamole / Placebo | Clopidogrel / Telmisartan | Clopidogrel / Placebo | Total
Number analyzed (Participants) | 5086 | 5095 | 5060 | 5091 | 20332
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (8.5) | 66.2 (8.6) | 66.2 (8.6) | 66.2 (8.5) | 66.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1802 | 1851 | 1817 | 1840 | 7310.0
  Male | 3284 | 3244 | 3243 | 3251 | 13022.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With First Recurrent Stroke of Any Type, Fatal or Nonfatal (Antiplatelet Comparison Only)
Time Frame: time since randomization; follow-up period is 1.5 to 4.4 years
Population: Patients were analyzed as randomized and were included in the analysis until final patient contact regardless of whether they were still on treatment.
Measure: Number; unit: Participants
Groups:
- Aspirin + Extended Release Dipyridamole: Consists of patients in the two treatment groups: ASA+ERDP + telmisartan and ASA+ERDP + placebo
- Clopidogrel: Consists of patients in the two treatment groups: Clopidogrel + telmisartan and Clopidogrel + placebo
Arm/Group | Aspirin + Extended Release Dipyridamole | Clopidogrel
Number analyzed (Participants) | 10181 | 10151
Participants | 916 | 898
Statistical Analysis 1: Comparison: Aspirin + Extended Release Dipyridamole vs Clopidogrel; ASA+ER-DP vs clopidogrel; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin of 1.075; p = 0.7830, Cox Proportional Hazard model; Cox proportional hazards model with age, baseline diabetes status, baseline ACE-I use, and baseline modified Rankin score as covariates; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.92 to 1.11]

2. Secondary Outcome: Composite Outcome of Stroke, Myocardial Infarction (MI), or Vascular Death (Antiplatelet Comparison Only)
Description: Number of patients with any of stroke, myocardial infarction, vascular death
Time Frame: time since randomization; follow-up period is 1.5 to 4.4 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Aspirin + Extended Release Dipyridamole | Clopidogrel
Number analyzed (Participants) | 10181 | 10151
Participants | 1333 | 1333
Statistical Analysis 1: Comparison: Aspirin + Extended Release Dipyridamole vs Clopidogrel; ASA+ER-DP vs Clopidogrel; Test type: Superiority or Other; p = 0.8292, Cox Proportional Hazard model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.92 to 1.07]

3. Secondary Outcome: Composite Outcome of Stroke, Myocardial Infarction, Vascular Death, or New or Worsening Congestive Heart Failure (CHF) (Telmisartan vs. Placebo Only)
Description: Number of patients with any of stroke, myocardial infarction, vascular death, or new or worsening congestive heart failure
Time Frame: time since randomization; follow-up period is 1.5 to 4.4 years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Telmisartan: Consists of patients in the two treatment groups: ASA+ERDP + telmisartan and Clopidogrel + telmisartan
- Placebo: Consists of patients in the two treatment groups: ASA+ERDP + placebo and Clopidogrel + placebo
Arm/Group | Telmisartan | Placebo
Number analyzed (Participants) | 10146 | 10186
Participants | 1367 | 1463
Statistical Analysis 1: Comparison: Telmisartan vs Placebo; Telmisartan vs Placebo; Test type: Superiority or Other; p = 0.1073, Cox Proportional Hazard model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.87 to 1.01]

4. Secondary Outcome: Number of Patients With New Onset of Diabetes (Telmisartan vs. Placebo Only)
Time Frame: Randomization to final patient contact
Population: Patients who did not have diabetes mellitus at baseline were analyzed as randomized and were included in the analysis until final patient contact regardless of whether they were still on treatment.
Measure: Number; unit: Participants
Arm/Group | Telmisartan | Placebo
Number analyzed (Participants) | 7306 | 7283
Participants | 125 | 151
Statistical Analysis 1: Comparison: Telmisartan vs Placebo; Telmisartan vs Placebo; Test type: Superiority or Other; p = 0.1007, Cox Proportional Hazard model; Cox proportional hazards model with age, baseline ACE-I use, and baseline modified Rankin score as covariates; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.04]

5. Primary Outcome: Number of Patients With First Recurrent Stroke of Any Type, Fatal or Nonfatal (Telmisartan vs. Placebo Only)
Time Frame: time since randomization; follow-up period is 1.5 to 4.4 years
Measure: Number; unit: Participants
Arm/Group | Telmisartan | Placebo
Number analyzed (Participants) | 10146 | 10186
Participants | 880 | 934
Statistical Analysis 1: Comparison: Telmisartan vs Placebo; Telmisartan vs placebo; Test type: Superiority or Other; p = 0.2312, Cox Proportional Hazard model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.86 to 1.04]

ADVERSE EVENTS:
Time Frame: From day of first dose until 28 days after last dose
Description: Treated Set of patients is used for Serious Adverse Events and Other Adverse Events analysis of Headache leading to permanent discontinuation. Randomized Set of patients is used for Dizziness assessed at Day 7 and Headache assessed at Day 7.
Arm/Group | Aspirin + Extended Release Dipyridamole / Telmisartan | Aspirin + Extended Release Dipyridamole / Placebo | Clopidogrel / Telmisartan | Clopidogrel / Placebo
Serious Adverse Events (participants affected / at risk) | 1145 | 1124 | 1225 | 1163
Other Adverse Events (participants affected / at risk) | 1856 | 1810 | 866 | 810
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Aspirin + Extended Release Dipyridamole / Telmisartan | Aspirin + Extended Release Dipyridamole / Placebo | Clopidogrel / Telmisartan | Clopidogrel / Placebo
Agranulocytosis (Blood and lymphatic system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Anaemia (Blood and lymphatic system disorders) | 21/5013 | 25/5024 | 21/5000 | 10/5023
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0/5013 | 2/5024 | 1/5000 | 0/5023
Aplastic anaemia (Blood and lymphatic system disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Eosinophilia (Blood and lymphatic system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Febrile neutropenia (Blood and lymphatic system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Haemolytic anaemia (Blood and lymphatic system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1/5013 | 0/5024 | 3/5000 | 1/5023
Leukocytosis (Blood and lymphatic system disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Leukopenia (Blood and lymphatic system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Lymphadenopathy (Blood and lymphatic system disorders) | 0/5013 | 0/5024 | 3/5000 | 0/5023
Microcytic anaemia (Blood and lymphatic system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1/5013 | 1/5024 | 2/5000 | 0/5023
Pancytopenia (Blood and lymphatic system disorders) | 5/5013 | 0/5024 | 1/5000 | 2/5023
Polycythaemia (Blood and lymphatic system disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Splenic infarction (Blood and lymphatic system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Thrombocythaemia (Blood and lymphatic system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Thrombocytopenia (Blood and lymphatic system disorders) | 1/5013 | 1/5024 | 0/5000 | 3/5023
AV dissociation (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Acute coronary syndrome (Cardiac disorders) | 3/5013 | 3/5024 | 3/5000 | 2/5023
Adams-Stokes syndrome (Cardiac disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Angina pectoris (Cardiac disorders) | 25/5013 | 18/5024 | 25/5000 | 20/5023
Angina unstable (Cardiac disorders) | 41/5013 | 47/5024 | 46/5000 | 30/5023
Aortic valve incompetence (Cardiac disorders) | 0/5013 | 2/5024 | 1/5000 | 1/5023
Aortic valve stenosis (Cardiac disorders) | 4/5013 | 0/5024 | 3/5000 | 1/5023
Arrhythmia (Cardiac disorders) | 3/5013 | 8/5024 | 5/5000 | 4/5023
Arrhythmia supraventricular (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Arteriosclerosis coronary artery (Cardiac disorders) | 1/5013 | 2/5024 | 2/5000 | 1/5023
Atrial fibrillation (Cardiac disorders) | 42/5013 | 38/5024 | 54/5000 | 47/5023
Atrial flutter (Cardiac disorders) | 2/5013 | 3/5024 | 4/5000 | 1/5023
Atrial tachycardia (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Atrioventricular block (Cardiac disorders) | 0/5013 | 1/5024 | 1/5000 | 2/5023
Atrioventricular block complete (Cardiac disorders) | 4/5013 | 3/5024 | 1/5000 | 4/5023
Atrioventricular block first degree (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Atrioventricular block second degree (Cardiac disorders) | 0/5013 | 0/5024 | 1/5000 | 3/5023
Bradyarrhythmia (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Bradycardia (Cardiac disorders) | 8/5013 | 4/5024 | 4/5000 | 8/5023
Cardiac aneurysm (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Cardiac arrest (Cardiac disorders) | 14/5013 | 5/5024 | 19/5000 | 8/5023
Cardiac disorder (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cardiac failure (Cardiac disorders) | 3/5013 | 5/5024 | 1/5000 | 2/5023
Cardiac failure acute (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 2/5023
Cardiac failure congestive (Cardiac disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Cardiac fibrillation (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cardiac hypertrophy (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Cardiac tamponade (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Cardiac valve disease (Cardiac disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Cardio-respiratory arrest (Cardiac disorders) | 2/5013 | 9/5024 | 5/5000 | 7/5023
Cardiogenic shock (Cardiac disorders) | 1/5013 | 0/5024 | 3/5000 | 0/5023
Cardiomyopathy (Cardiac disorders) | 1/5013 | 1/5024 | 1/5000 | 3/5023
Cardiopulmonary failure (Cardiac disorders) | 0/5013 | 0/5024 | 3/5000 | 1/5023
Cardiovascular disorder (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Conduction disorder (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Congestive cardiomyopathy (Cardiac disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Cor pulmonale (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Cor pulmonale acute (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Coronary artery disease (Cardiac disorders) | 14/5013 | 33/5024 | 21/5000 | 31/5023
Coronary artery dissection (Cardiac disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Coronary artery occlusion (Cardiac disorders) | 1/5013 | 0/5024 | 2/5000 | 2/5023
Coronary artery restenosis (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Coronary artery stenosis (Cardiac disorders) | 9/5013 | 4/5024 | 9/5000 | 5/5023
Electromechanical dissociation (Cardiac disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Extrasystoles (Cardiac disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Haemorrhage coronary artery (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hypertensive heart disease (Cardiac disorders) | 0/5013 | 1/5024 | 3/5000 | 0/5023
Hypertrophic cardiomyopathy (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
In-stent coronary artery restenosis (Cardiac disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Intracardiac thrombus (Cardiac disorders) | 2/5013 | 1/5024 | 0/5000 | 2/5023
Left ventricular dysfunction (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Left ventricular failure (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Left ventricular hypertrophy (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Mitral valve calcification (Cardiac disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Mitral valve incompetence (Cardiac disorders) | 2/5013 | 0/5024 | 2/5000 | 0/5023
Mitral valve prolapse (Cardiac disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Mitral valve stenosis (Cardiac disorders) | 0/5013 | 1/5024 | 2/5000 | 0/5023
Myocardial infarction (Cardiac disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Myocardial ischaemia (Cardiac disorders) | 4/5013 | 8/5024 | 2/5000 | 5/5023
Myopericarditis (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Palpitations (Cardiac disorders) | 3/5013 | 3/5024 | 5/5000 | 1/5023
Pericardial effusion (Cardiac disorders) | 0/5013 | 2/5024 | 2/5000 | 0/5023
Pericarditis (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Sick sinus syndrome (Cardiac disorders) | 3/5013 | 2/5024 | 3/5000 | 2/5023
Sinus arrest (Cardiac disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Sinus bradycardia (Cardiac disorders) | 1/5013 | 0/5024 | 1/5000 | 2/5023
Sinus tachycardia (Cardiac disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Supraventricular extrasystoles (Cardiac disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Supraventricular tachycardia (Cardiac disorders) | 5/5013 | 5/5024 | 3/5000 | 0/5023
Tachyarrhythmia (Cardiac disorders) | 1/5013 | 0/5024 | 3/5000 | 1/5023
Tachycardia (Cardiac disorders) | 0/5013 | 0/5024 | 3/5000 | 4/5023
Tachycardia paroxysmal (Cardiac disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Ventricular arrhythmia (Cardiac disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Ventricular extrasystoles (Cardiac disorders) | 2/5013 | 0/5024 | 3/5000 | 2/5023
Ventricular fibrillation (Cardiac disorders) | 1/5013 | 0/5024 | 3/5000 | 1/5023
Ventricular tachycardia (Cardiac disorders) | 0/5013 | 2/5024 | 3/5000 | 3/5023
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Atrial septal defect (Congenital, familial and genetic disorders) | 1/5013 | 2/5024 | 2/5000 | 3/5023
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Corneal dystrophy (Congenital, familial and genetic disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hydrocele (Congenital, familial and genetic disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Hypospadias (Congenital, familial and genetic disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Spondylolisthesis (Congenital, familial and genetic disorders) | 0/5013 | 3/5024 | 1/5000 | 0/5023
Conductive deafness (Ear and labyrinth disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Deafness (Ear and labyrinth disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Deafness unilateral (Ear and labyrinth disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Ear haemorrhage (Ear and labyrinth disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Ear pain (Ear and labyrinth disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Hypoacusis (Ear and labyrinth disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Meniere's disease (Ear and labyrinth disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Sudden hearing loss (Ear and labyrinth disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Tympanic membrane perforation (Ear and labyrinth disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Vertigo (Ear and labyrinth disorders) | 13/5013 | 12/5024 | 20/5000 | 10/5023
Vertigo labyrinthine (Ear and labyrinth disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Vertigo positional (Ear and labyrinth disorders) | 2/5013 | 2/5024 | 5/5000 | 2/5023
Vestibular disorder (Ear and labyrinth disorders) | 2/5013 | 2/5024 | 1/5000 | 2/5023
Vestibular neuronitis (Ear and labyrinth disorders) | 2/5013 | 3/5024 | 0/5000 | 0/5023
Basedow's disease (Endocrine disorders) | 0/5013 | 2/5024 | 0/5000 | 0/5023
Euthyroid sick syndrome (Endocrine disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Goitre (Endocrine disorders) | 6/5013 | 0/5024 | 1/5000 | 2/5023
Hyperaldosteronism (Endocrine disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hyperparathyroidism (Endocrine disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hyperthyroidism (Endocrine disorders) | 3/5013 | 2/5024 | 1/5000 | 1/5023
Hypothyroidism (Endocrine disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0/5013 | 0/5024 | 1/5000 | 2/5023
Parathyroid gland enlargement (Endocrine disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Thyrotoxic crisis (Endocrine disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Angle closure glaucoma (Eye disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cataract (Eye disorders) | 12/5013 | 15/5024 | 9/5000 | 8/5023
Dacryostenosis acquired (Eye disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Diabetic retinopathy (Eye disorders) | 1/5013 | 2/5024 | 1/5000 | 0/5023
Diplopia (Eye disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Eyelid ptosis (Eye disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Glaucoma (Eye disorders) | 2/5013 | 1/5024 | 2/5000 | 1/5023
Keratitis (Eye disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Maculopathy (Eye disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Open angle glaucoma (Eye disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Retinal detachment (Eye disorders) | 0/5013 | 2/5024 | 2/5000 | 2/5023
Retinal haemorrhage (Eye disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Retinal tear (Eye disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Retinal vein occlusion (Eye disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Strabismus (Eye disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Ulcerative keratitis (Eye disorders) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Uveitis (Eye disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Vision blurred (Eye disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Visual acuity reduced (Eye disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Visual disturbance (Eye disorders) | 0/5013 | 1/5024 | 2/5000 | 1/5023
Abdominal discomfort (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 2/5023
Abdominal distension (Gastrointestinal disorders) | 0/5013 | 0/5024 | 2/5000 | 2/5023
Abdominal hernia (Gastrointestinal disorders) | 2/5013 | 1/5024 | 0/5000 | 2/5023
Abdominal mass (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Abdominal pain (Gastrointestinal disorders) | 10/5013 | 12/5024 | 13/5000 | 7/5023
Abdominal pain lower (Gastrointestinal disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Abdominal pain upper (Gastrointestinal disorders) | 6/5013 | 2/5024 | 2/5000 | 6/5023
Abdominal strangulated hernia (Gastrointestinal disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Acute abdomen (Gastrointestinal disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Anal fissure (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Anal fistula (Gastrointestinal disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Anal prolapse (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Anal ulcer (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Aphagia (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Appendicitis perforated (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Ascites (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Barrett's oesophagus (Gastrointestinal disorders) | 1/5013 | 0/5024 | 1/5000 | 2/5023
Colitis (Gastrointestinal disorders) | 1/5013 | 0/5024 | 2/5000 | 2/5023
Colitis ischaemic (Gastrointestinal disorders) | 2/5013 | 2/5024 | 1/5000 | 1/5023
Colitis ulcerative (Gastrointestinal disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Colonic obstruction (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Colonic polyp (Gastrointestinal disorders) | 7/5013 | 6/5024 | 3/5000 | 2/5023
Constipation (Gastrointestinal disorders) | 3/5013 | 2/5024 | 1/5000 | 5/5023
Crohn's disease (Gastrointestinal disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Diabetic gastroparesis (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Diarrhoea (Gastrointestinal disorders) | 18/5013 | 18/5024 | 18/5000 | 10/5023
Diverticulum (Gastrointestinal disorders) | 2/5013 | 2/5024 | 1/5000 | 0/5023
Diverticulum intestinal (Gastrointestinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Duodenal ulcer (Gastrointestinal disorders) | 10/5013 | 4/5024 | 9/5000 | 12/5023
Duodenal ulcer perforation (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Duodenitis (Gastrointestinal disorders) | 4/5013 | 1/5024 | 0/5000 | 1/5023
Dyspepsia (Gastrointestinal disorders) | 2/5013 | 1/5024 | 0/5000 | 2/5023
Dysphagia (Gastrointestinal disorders) | 2/5013 | 3/5024 | 5/5000 | 4/5023
Enteritis (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Enterocolitis (Gastrointestinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Erosive oesophagitis (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Faecaloma (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Femoral hernia (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Femoral hernia, obstructive (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Gastric polyps (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Gastric ulcer (Gastrointestinal disorders) | 13/5013 | 8/5024 | 10/5000 | 8/5023
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Gastric ulcer perforation (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Gastritis (Gastrointestinal disorders) | 7/5013 | 8/5024 | 5/5000 | 7/5023
Gastritis erosive (Gastrointestinal disorders) | 4/5013 | 4/5024 | 2/5000 | 1/5023
Gastroduodenal ulcer (Gastrointestinal disorders) | 2/5013 | 2/5024 | 0/5000 | 2/5023
Gastroduodenitis (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Gastrointestinal disorder (Gastrointestinal disorders) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Gastrointestinal necrosis (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/5013 | 4/5024 | 5/5000 | 2/5023
Gastrooesophagitis (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Gingivitis (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Haemorrhoids (Gastrointestinal disorders) | 1/5013 | 2/5024 | 1/5000 | 1/5023
Hiatus hernia (Gastrointestinal disorders) | 2/5013 | 1/5024 | 2/5000 | 0/5023
Ileitis (Gastrointestinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Ileus (Gastrointestinal disorders) | 2/5013 | 1/5024 | 3/5000 | 1/5023
Ileus paralytic (Gastrointestinal disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Inguinal hernia (Gastrointestinal disorders) | 6/5013 | 17/5024 | 10/5000 | 17/5023
Inguinal hernia strangulated (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Intestinal ischaemia (Gastrointestinal disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Intestinal obstruction (Gastrointestinal disorders) | 4/5013 | 3/5024 | 4/5000 | 6/5023
Intestinal perforation (Gastrointestinal disorders) | 0/5013 | 2/5024 | 2/5000 | 0/5023
Irritable bowel syndrome (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Mechanical ileus (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Megacolon (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Mesenteric arteriosclerosis (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Mesenteric artery stenosis (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Mouth ulceration (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Nausea (Gastrointestinal disorders) | 13/5013 | 10/5024 | 8/5000 | 4/5023
Oedematous pancreatitis (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Oesophageal polyp (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Oesophageal stenosis (Gastrointestinal disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Oesophageal ulcer (Gastrointestinal disorders) | 0/5013 | 1/5024 | 3/5000 | 0/5023
Oesophagitis (Gastrointestinal disorders) | 2/5013 | 2/5024 | 0/5000 | 2/5023
Oesophagitis ulcerative (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Oral disorder (Gastrointestinal disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Oral mucosal blistering (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Pancreatic mass (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pancreatic necrosis (Gastrointestinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Pancreatitis (Gastrointestinal disorders) | 6/5013 | 5/5024 | 4/5000 | 7/5023
Pancreatitis acute (Gastrointestinal disorders) | 2/5013 | 3/5024 | 7/5000 | 1/5023
Pancreatitis chronic (Gastrointestinal disorders) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Paraesthesia oral (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Peptic ulcer (Gastrointestinal disorders) | 1/5013 | 3/5024 | 0/5000 | 1/5023
Periodontitis (Gastrointestinal disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Peritonitis (Gastrointestinal disorders) | 1/5013 | 2/5024 | 1/5000 | 1/5023
Proctalgia (Gastrointestinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Proctitis (Gastrointestinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Proctocolitis (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Rectal polyp (Gastrointestinal disorders) | 2/5013 | 0/5024 | 2/5000 | 0/5023
Rectal prolapse (Gastrointestinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Rectal stenosis (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Rectal ulcer (Gastrointestinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Reflux oesophagitis (Gastrointestinal disorders) | 1/5013 | 2/5024 | 2/5000 | 2/5023
Small intestinal obstruction (Gastrointestinal disorders) | 7/5013 | 2/5024 | 1/5000 | 3/5023
Stomach mass (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Tongue oedema (Gastrointestinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Tooth disorder (Gastrointestinal disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Umbilical hernia (Gastrointestinal disorders) | 1/5013 | 2/5024 | 2/5000 | 0/5023
Varices oesophageal (Gastrointestinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Volvulus (Gastrointestinal disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Vomiting (Gastrointestinal disorders) | 23/5013 | 18/5024 | 13/5000 | 15/5023
Adverse drug reaction (General disorders) | 0/5013 | 7/5024 | 4/5000 | 4/5023
Asthenia (General disorders) | 5/5013 | 7/5024 | 11/5000 | 7/5023
Calcinosis (General disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cardiac death (General disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Catheter site haemorrhage (General disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Chest discomfort (General disorders) | 4/5013 | 1/5024 | 3/5000 | 2/5023
Chest pain (General disorders) | 44/5013 | 33/5024 | 21/5000 | 30/5023
Chills (General disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Death (General disorders) | 39/5013 | 37/5024 | 39/5000 | 34/5023
Drowning (General disorders) | 3/5013 | 0/5024 | 0/5000 | 1/5023
Drug withdrawal syndrome (General disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Dysplasia (General disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Effusion (General disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Face oedema (General disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Facial pain (General disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Fatigue (General disorders) | 4/5013 | 4/5024 | 3/5000 | 1/5023
Feeling abnormal (General disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Fibrosis (General disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Gait disturbance (General disorders) | 5/5013 | 3/5024 | 5/5000 | 1/5023
General physical health deterioration (General disorders) | 3/5013 | 3/5024 | 1/5000 | 1/5023
Generalised oedema (General disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Granuloma (General disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hernia (General disorders) | 0/5013 | 0/5024 | 3/5000 | 0/5023
Hyperthermia (General disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Hyperthermia malignant (General disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Hypothermia (General disorders) | 0/5013 | 2/5024 | 0/5000 | 0/5023
Impaired healing (General disorders) | 1/5013 | 0/5024 | 1/5000 | 4/5023
Influenza like illness (General disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Malaise (General disorders) | 5/5013 | 2/5024 | 1/5000 | 3/5023
Multi-organ disorder (General disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Multi-organ failure (General disorders) | 1/5013 | 2/5024 | 3/5000 | 1/5023
Non-cardiac chest pain (General disorders) | 3/5013 | 4/5024 | 1/5000 | 1/5023
Oedema (General disorders) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Oedema peripheral (General disorders) | 4/5013 | 1/5024 | 1/5000 | 3/5023
Pain (General disorders) | 0/5013 | 0/5024 | 2/5000 | 4/5023
Polyp (General disorders) | 2/5013 | 2/5024 | 0/5000 | 0/5023
Pyrexia (General disorders) | 15/5013 | 11/5024 | 12/5000 | 12/5023
Sudden cardiac death (General disorders) | 4/5013 | 0/5024 | 1/5000 | 1/5023
Sudden death (General disorders) | 5/5013 | 3/5024 | 4/5000 | 5/5023
Systemic inflammatory response syndrome (General disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Tenderness (General disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Ulcer (General disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Vestibulitis (General disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Acute hepatic failure (Hepatobiliary disorders) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Bile duct obstruction (Hepatobiliary disorders) | 0/5013 | 0/5024 | 1/5000 | 2/5023
Bile duct stone (Hepatobiliary disorders) | 3/5013 | 4/5024 | 3/5000 | 3/5023
Biliary colic (Hepatobiliary disorders) | 0/5013 | 1/5024 | 0/5000 | 2/5023
Cholangitis (Hepatobiliary disorders) | 4/5013 | 2/5024 | 1/5000 | 4/5023
Cholangitis acute (Hepatobiliary disorders) | 2/5013 | 1/5024 | 0/5000 | 2/5023
Cholecystitis (Hepatobiliary disorders) | 5/5013 | 5/5024 | 3/5000 | 6/5023
Cholecystitis acute (Hepatobiliary disorders) | 2/5013 | 10/5024 | 9/5000 | 5/5023
Cholecystitis chronic (Hepatobiliary disorders) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Cholelithiasis (Hepatobiliary disorders) | 10/5013 | 8/5024 | 9/5000 | 9/5023
Gallbladder disorder (Hepatobiliary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Gallbladder necrosis (Hepatobiliary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Gallbladder pain (Hepatobiliary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Gallbladder polyp (Hepatobiliary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hepatic cirrhosis (Hepatobiliary disorders) | 0/5013 | 2/5024 | 0/5000 | 2/5023
Hepatic failure (Hepatobiliary disorders) | 0/5013 | 1/5024 | 0/5000 | 3/5023
Hepatic function abnormal (Hepatobiliary disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Hepatic steatosis (Hepatobiliary disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Hepatitis (Hepatobiliary disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Hepatitis acute (Hepatobiliary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Hepatitis toxic (Hepatobiliary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hepatomegaly (Hepatobiliary disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Hyperbilirubinaemia (Hepatobiliary disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Jaundice (Hepatobiliary disorders) | 2/5013 | 0/5024 | 1/5000 | 0/5023
Jaundice cholestatic (Hepatobiliary disorders) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Liver disorder (Hepatobiliary disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Allergic oedema (Immune system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Anaphylactic reaction (Immune system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Anaphylactic shock (Immune system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Drug hypersensitivity (Immune system disorders) | 0/5013 | 0/5024 | 1/5000 | 2/5023
Food allergy (Immune system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Hypersensitivity (Immune system disorders) | 0/5013 | 3/5024 | 1/5000 | 5/5023
Sarcoidosis (Immune system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Abdominal abscess (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Abdominal wall abscess (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Abscess (Infections and infestations) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Abscess intestinal (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Abscess limb (Infections and infestations) | 1/5013 | 0/5024 | 2/5000 | 2/5023
Abscess oral (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Acute tonsillitis (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Anal abscess (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Anogenital warts (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Appendicitis (Infections and infestations) | 5/5013 | 5/5024 | 5/5000 | 8/5023
Arthritis bacterial (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Arthritis infective (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Aspergillosis (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Bacteraemia (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Bacterial sepsis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Bone tuberculosis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Borrelia infection (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Breast abscess (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Bronchiectasis (Infections and infestations) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Bronchitis (Infections and infestations) | 11/5013 | 5/5024 | 6/5000 | 7/5023
Bronchopneumonia (Infections and infestations) | 4/5013 | 2/5024 | 2/5000 | 5/5023
Bronchopulmonary aspergillosis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Burn infection (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Bursitis infective (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Campylobacter intestinal infection (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Carbuncle (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Catheter related infection (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Catheter sepsis (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Catheter site infection (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Cellulitis (Infections and infestations) | 9/5013 | 5/5024 | 11/5000 | 8/5023
Cellulitis pharyngeal (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cellulitis staphylococcal (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cholecystitis infective (Infections and infestations) | 0/5013 | 2/5024 | 1/5000 | 1/5023
Chronic sinusitis (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Clostridial infection (Infections and infestations) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Clostridium difficile colitis (Infections and infestations) | 2/5013 | 1/5024 | 1/5000 | 0/5023
Cystitis (Infections and infestations) | 2/5013 | 1/5024 | 6/5000 | 1/5023
Dengue fever (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Device related infection (Infections and infestations) | 0/5013 | 1/5024 | 2/5000 | 0/5023
Diabetic gangrene (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Diarrhoea infectious (Infections and infestations) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Disseminated tuberculosis (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Diverticulitis (Infections and infestations) | 3/5013 | 5/5024 | 5/5000 | 1/5023
Dysentery (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Empyema (Infections and infestations) | 2/5013 | 0/5024 | 0/5000 | 1/5023
Encephalitis viral (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Endocarditis (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Endocarditis bacterial (Infections and infestations) | 0/5013 | 1/5024 | 2/5000 | 0/5023
Endocarditis enterococcal (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Endometritis (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Enteritis infectious (Infections and infestations) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Enterococcal sepsis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Epidemic vomiting syndrome (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Epiglottitis (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Erysipelas (Infections and infestations) | 1/5013 | 1/5024 | 1/5000 | 4/5023
Escherichia infection (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Escherichia sepsis (Infections and infestations) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Escherichia urinary tract infection (Infections and infestations) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Febrile infection (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Fungal infection (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Gangrene (Infections and infestations) | 2/5013 | 1/5024 | 1/5000 | 4/5023
Gastritis viral (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Gastroenteritis (Infections and infestations) | 17/5013 | 8/5024 | 14/5000 | 10/5023
Gastroenteritis viral (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Gastrointestinal infection (Infections and infestations) | 2/5013 | 0/5024 | 2/5000 | 0/5023
Genitourinary tract infection (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Graft infection (Infections and infestations) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Helicobacter gastritis (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Hepatitis A (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hepatitis B (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hepatitis C (Infections and infestations) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Hepatitis E (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Hepatitis viral (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Herpes zoster (Infections and infestations) | 1/5013 | 1/5024 | 3/5000 | 4/5023
Incision site abscess (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Infected epidermal cyst (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Infected skin ulcer (Infections and infestations) | 0/5013 | 1/5024 | 3/5000 | 0/5023
Infection (Infections and infestations) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1/5013 | 0/5024 | 5/5000 | 1/5023
Influenza (Infections and infestations) | 0/5013 | 1/5024 | 2/5000 | 1/5023
Joint abscess (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Kidney infection (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Klebsiella bacteraemia (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Klebsiella infection (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Labyrinthitis (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Liver abscess (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lobar pneumonia (Infections and infestations) | 2/5013 | 3/5024 | 5/5000 | 4/5023
Localised infection (Infections and infestations) | 5/5013 | 1/5024 | 2/5000 | 5/5023
Lower respiratory tract infection (Infections and infestations) | 4/5013 | 2/5024 | 5/5000 | 4/5023
Lung abscess (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lung infection (Infections and infestations) | 6/5013 | 4/5024 | 3/5000 | 3/5023
Lymph node tuberculosis (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Malaria (Infections and infestations) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Mastoiditis (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Meningitis (Infections and infestations) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Meningitis bacterial (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Meningitis tuberculous (Infections and infestations) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Nasopharyngitis (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Necrotising fasciitis (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Oropharyngeal candidiasis (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Osteomyelitis (Infections and infestations) | 3/5013 | 1/5024 | 1/5000 | 1/5023
Osteomyelitis acute (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Osteomyelitis chronic (Infections and infestations) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Otitis externa (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Otitis media (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Otitis media acute (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Paronychia (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Parotitis (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Perianal abscess (Infections and infestations) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Pericarditis tuberculous (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Perineal abscess (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Perinephric abscess (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Perirectal abscess (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Peritonsillar abscess (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Plasmodium falciparum infection (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Pneumococcal bacteraemia (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Pneumonia (Infections and infestations) | 62/5013 | 60/5024 | 72/5000 | 73/5023
Pneumonia pneumococcal (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Pneumonia primary atypical (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pneumonia streptococcal (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Post procedural infection (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Postoperative wound infection (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pseudomembranous colitis (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Pulmonary sepsis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pulmonary tuberculosis (Infections and infestations) | 3/5013 | 1/5024 | 1/5000 | 2/5023
Purulence (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Purulent discharge (Infections and infestations) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Pyelonephritis (Infections and infestations) | 1/5013 | 3/5024 | 5/5000 | 3/5023
Pyelonephritis acute (Infections and infestations) | 1/5013 | 4/5024 | 1/5000 | 0/5023
Pyelonephritis chronic (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Pyothorax (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Rectal abscess (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Respiratory tract infection (Infections and infestations) | 3/5013 | 2/5024 | 3/5000 | 3/5023
Respiratory tract infection viral (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Salmonella sepsis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Salmonellosis (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Scrotal abscess (Infections and infestations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Sepsis (Infections and infestations) | 17/5013 | 11/5024 | 17/5000 | 14/5023
Septic embolus (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Septic shock (Infections and infestations) | 3/5013 | 6/5024 | 7/5000 | 2/5023
Sialoadenitis (Infections and infestations) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Sinusitis (Infections and infestations) | 2/5013 | 4/5024 | 0/5000 | 0/5023
Staphylococcal infection (Infections and infestations) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Stitch abscess (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Streptococcal sepsis (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Subcutaneous abscess (Infections and infestations) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Sweat gland infection (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Tonsillitis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Tooth infection (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Toxic shock syndrome (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Tracheobronchitis (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Tuberculosis (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Tuberculous pleurisy (Infections and infestations) | 0/5013 | 2/5024 | 0/5000 | 0/5023
Typhoid fever (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Upper respiratory tract infection (Infections and infestations) | 3/5013 | 5/5024 | 3/5000 | 1/5023
Urinary bladder abscess (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Urinary tract infection (Infections and infestations) | 32/5013 | 22/5024 | 40/5000 | 38/5023
Urinary tract infection enterococcal (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Urosepsis (Infections and infestations) | 2/5013 | 3/5024 | 9/5000 | 6/5023
Viral infection (Infections and infestations) | 1/5013 | 3/5024 | 2/5000 | 1/5023
Viral myocarditis (Infections and infestations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Viral pharyngitis (Infections and infestations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Viral upper respiratory tract infection (Infections and infestations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
West Nile viral infection (Infections and infestations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Wound infection (Infections and infestations) | 1/5013 | 2/5024 | 1/5000 | 2/5023
Accident (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Accident at work (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Accidental overdose (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Acetabulum fracture (Injury, poisoning and procedural complications) | 0/5013 | 2/5024 | 1/5000 | 1/5023
Alcohol poisoning (Injury, poisoning and procedural complications) | 3/5013 | 0/5024 | 1/5000 | 4/5023
Anaemia postoperative (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Animal bite (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Ankle fracture (Injury, poisoning and procedural complications) | 3/5013 | 4/5024 | 4/5000 | 1/5023
Arthropod bite (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Avulsion fracture (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Back injury (Injury, poisoning and procedural complications) | 0/5013 | 2/5024 | 2/5000 | 1/5023
Brain contusion (Injury, poisoning and procedural complications) | 3/5013 | 0/5024 | 0/5000 | 2/5023
Burns second degree (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Burns third degree (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2/5013 | 1/5024 | 1/5000 | 1/5023
Chemical poisoning (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Clavicle fracture (Injury, poisoning and procedural complications) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Collapse of lung (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Comminuted fracture (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Compression fracture (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Concussion (Injury, poisoning and procedural complications) | 2/5013 | 3/5024 | 0/5000 | 4/5023
Contusion (Injury, poisoning and procedural complications) | 3/5013 | 3/5024 | 1/5000 | 4/5023
Device failure (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Drug toxicity (Injury, poisoning and procedural complications) | 2/5013 | 3/5024 | 0/5000 | 2/5023
Eschar (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Excoriation (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Extradural haematoma (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Eye injury (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 2/5023
Eye penetration (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Face injury (Injury, poisoning and procedural complications) | 0/5013 | 2/5024 | 1/5000 | 1/5023
Facial bones fracture (Injury, poisoning and procedural complications) | 2/5013 | 2/5024 | 0/5000 | 2/5023
Fall (Injury, poisoning and procedural complications) | 39/5013 | 53/5024 | 40/5000 | 49/5023
Femoral neck fracture (Injury, poisoning and procedural complications) | 9/5013 | 13/5024 | 12/5000 | 9/5023
Femur fracture (Injury, poisoning and procedural complications) | 11/5013 | 12/5024 | 13/5000 | 12/5023
Fibula fracture (Injury, poisoning and procedural complications) | 2/5013 | 0/5024 | 2/5000 | 0/5023
Foot fracture (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 2/5000 | 1/5023
Forearm fracture (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Foreign body in eye (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Foreign body trauma (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Fracture (Injury, poisoning and procedural complications) | 4/5013 | 1/5024 | 1/5000 | 2/5023
Fracture displacement (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Fractured coccyx (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hand fracture (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 3/5023
Head injury (Injury, poisoning and procedural complications) | 9/5013 | 9/5024 | 9/5000 | 12/5023
Heat exhaustion (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Heat stroke (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Hip fracture (Injury, poisoning and procedural complications) | 14/5013 | 15/5024 | 12/5000 | 12/5023
Humerus fracture (Injury, poisoning and procedural complications) | 4/5013 | 5/5024 | 10/5000 | 5/5023
Ilium fracture (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Incisional hernia (Injury, poisoning and procedural complications) | 2/5013 | 1/5024 | 2/5000 | 0/5023
Injury (Injury, poisoning and procedural complications) | 3/5013 | 2/5024 | 3/5000 | 3/5023
Jaw fracture (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Joint dislocation (Injury, poisoning and procedural complications) | 3/5013 | 2/5024 | 5/5000 | 2/5023
Joint injury (Injury, poisoning and procedural complications) | 0/5013 | 2/5024 | 2/5000 | 1/5023
Joint sprain (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Limb injury (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Lower limb fracture (Injury, poisoning and procedural complications) | 0/5013 | 4/5024 | 1/5000 | 0/5023
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1/5013 | 2/5024 | 0/5000 | 3/5023
Medical device pain (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Medication error (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Meniscus lesion (Injury, poisoning and procedural complications) | 1/5013 | 4/5024 | 0/5000 | 1/5023
Multiple drug overdose (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Multiple fractures (Injury, poisoning and procedural complications) | 1/5013 | 1/5024 | 2/5000 | 1/5023
Multiple injuries (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 2/5000 | 2/5023
Muscle injury (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Muscle strain (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Neck injury (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 2/5000 | 1/5023
Nerve injury (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Open wound (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Overdose (Injury, poisoning and procedural complications) | 2/5013 | 0/5024 | 2/5000 | 0/5023
Pacemaker complication (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Patella fracture (Injury, poisoning and procedural complications) | 1/5013 | 1/5024 | 3/5000 | 0/5023
Pelvic fracture (Injury, poisoning and procedural complications) | 5/5013 | 2/5024 | 3/5000 | 4/5023
Periorbital haematoma (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Post procedural fistula (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Postoperative fever (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Postoperative ileus (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Procedural pain (Injury, poisoning and procedural complications) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Procedural site reaction (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pubic rami fracture (Injury, poisoning and procedural complications) | 3/5013 | 0/5024 | 0/5000 | 0/5023
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Radius fracture (Injury, poisoning and procedural complications) | 3/5013 | 0/5024 | 1/5000 | 2/5023
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Rib fracture (Injury, poisoning and procedural complications) | 3/5013 | 5/5024 | 4/5000 | 4/5023
Road traffic accident (Injury, poisoning and procedural complications) | 10/5013 | 9/5024 | 7/5000 | 12/5023
Scapula fracture (Injury, poisoning and procedural complications) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Scratch (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Shunt aneurysm (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Skeletal injury (Injury, poisoning and procedural complications) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Skin laceration (Injury, poisoning and procedural complications) | 4/5013 | 2/5024 | 4/5000 | 1/5023
Skull fracture (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Snake bite (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Spinal compression fracture (Injury, poisoning and procedural complications) | 5/5013 | 1/5024 | 6/5000 | 6/5023
Spinal cord injury (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Spinal fracture (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Splenic rupture (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Sports injury (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Stent occlusion (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Sternal fracture (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Subdural haematoma (Injury, poisoning and procedural complications) | 3/5013 | 3/5024 | 4/5000 | 8/5023
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2/5013 | 1/5024 | 3/5000 | 2/5023
Synovial rupture (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Tendon rupture (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Thermal burn (Injury, poisoning and procedural complications) | 2/5013 | 0/5024 | 1/5000 | 1/5023
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1/5013 | 1/5024 | 1/5000 | 2/5023
Tibia fracture (Injury, poisoning and procedural complications) | 2/5013 | 1/5024 | 2/5000 | 1/5023
Traumatic arthritis (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Traumatic brain injury (Injury, poisoning and procedural complications) | 2/5013 | 1/5024 | 0/5000 | 2/5023
Traumatic fracture (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Traumatic ulcer (Injury, poisoning and procedural complications) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Ulna fracture (Injury, poisoning and procedural complications) | 1/5013 | 2/5024 | 2/5000 | 2/5023
Upper limb fracture (Injury, poisoning and procedural complications) | 7/5013 | 1/5024 | 5/5000 | 3/5023
Vaccination complication (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Wound (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Wound dehiscence (Injury, poisoning and procedural complications) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Wrist fracture (Injury, poisoning and procedural complications) | 2/5013 | 3/5024 | 2/5000 | 1/5023
Acid base balance abnormal (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Alanine aminotransferase increased (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Allergy test (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Arteriogram coronary (Investigations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Aspartate aminotransferase increased (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Aspiration bronchial (Investigations) | 1/5013 | 1/5024 | 3/5000 | 0/5023
Biopsy lymph gland (Investigations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Blood creatine phosphokinase increased (Investigations) | 0/5013 | 0/5024 | 0/5000 | 3/5023
Blood creatinine increased (Investigations) | 1/5013 | 4/5024 | 6/5000 | 3/5023
Blood glucose abnormal (Investigations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Blood glucose decreased (Investigations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Blood glucose increased (Investigations) | 0/5013 | 3/5024 | 2/5000 | 0/5023
Blood lactate dehydrogenase increased (Investigations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Blood potassium decreased (Investigations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Blood potassium increased (Investigations) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Blood pressure decreased (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Blood pressure increased (Investigations) | 4/5013 | 3/5024 | 2/5000 | 1/5023
Blood pressure systolic increased (Investigations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Blood sodium decreased (Investigations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Blood test abnormal (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Blood urea increased (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Body temperature increased (Investigations) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Cardiac enzymes increased (Investigations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Creatinine renal clearance decreased (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Endoscopic retrograde cholangiopancreatography (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Haematocrit decreased (Investigations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Haemoglobin decreased (Investigations) | 3/5013 | 1/5024 | 1/5000 | 2/5023
Heart rate decreased (Investigations) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Heart rate irregular (Investigations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hepatic enzyme increased (Investigations) | 2/5013 | 0/5024 | 1/5000 | 1/5023
International normalised ratio increased (Investigations) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Liver function test abnormal (Investigations) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Myoglobin blood increased (Investigations) | 0/5013 | 0/5024 | 0/5000 | 1/5023
QRS axis abnormal (Investigations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Renal function test abnormal (Investigations) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Transaminases increased (Investigations) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Troponin increased (Investigations) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Urine output decreased (Investigations) | 0/5013 | 2/5024 | 0/5000 | 1/5023
Weight decreased (Investigations) | 4/5013 | 1/5024 | 1/5000 | 3/5023
Anorexia (Metabolism and nutrition disorders) | 2/5013 | 3/5024 | 1/5000 | 1/5023
Cachexia (Metabolism and nutrition disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Decreased appetite (Metabolism and nutrition disorders) | 2/5013 | 0/5024 | 1/5000 | 1/5023
Dehydration (Metabolism and nutrition disorders) | 27/5013 | 22/5024 | 12/5000 | 7/5023
Diabetes mellitus (Metabolism and nutrition disorders) | 3/5013 | 6/5024 | 4/5000 | 3/5023
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 6/5013 | 6/5024 | 6/5000 | 6/5023
Diabetic complication (Metabolism and nutrition disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Diabetic foot (Metabolism and nutrition disorders) | 2/5013 | 4/5024 | 2/5000 | 2/5023
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3/5013 | 1/5024 | 2/5000 | 0/5023
Electrolyte imbalance (Metabolism and nutrition disorders) | 2/5013 | 0/5024 | 1/5000 | 0/5023
Failure to thrive (Metabolism and nutrition disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Fluid overload (Metabolism and nutrition disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Gout (Metabolism and nutrition disorders) | 1/5013 | 2/5024 | 1/5000 | 4/5023
Hypercalcaemia (Metabolism and nutrition disorders) | 1/5013 | 0/5024 | 1/5000 | 3/5023
Hyperglycaemia (Metabolism and nutrition disorders) | 2/5013 | 2/5024 | 8/5000 | 4/5023
Hyperkalaemia (Metabolism and nutrition disorders) | 8/5013 | 0/5024 | 5/5000 | 4/5023
Hyperuricaemia (Metabolism and nutrition disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Hypochloraemia (Metabolism and nutrition disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Hypoglycaemia (Metabolism and nutrition disorders) | 13/5013 | 11/5024 | 18/5000 | 10/5023
Hypokalaemia (Metabolism and nutrition disorders) | 3/5013 | 5/5024 | 4/5000 | 7/5023
Hyponatraemia (Metabolism and nutrition disorders) | 13/5013 | 18/5024 | 19/5000 | 11/5023
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Hypovolaemia (Metabolism and nutrition disorders) | 0/5013 | 2/5024 | 0/5000 | 1/5023
Ketosis (Metabolism and nutrition disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Lactic acidosis (Metabolism and nutrition disorders) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Malnutrition (Metabolism and nutrition disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Metabolic acidosis (Metabolism and nutrition disorders) | 2/5013 | 1/5024 | 1/5000 | 1/5023
Metabolic alkalosis (Metabolism and nutrition disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Obesity (Metabolism and nutrition disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Oral intake reduced (Metabolism and nutrition disorders) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Overweight (Metabolism and nutrition disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 3/5013 | 0/5024 | 0/5000 | 0/5023
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/5013 | 4/5024 | 4/5000 | 7/5023
Arthritis (Musculoskeletal and connective tissue disorders) | 0/5013 | 2/5024 | 4/5000 | 0/5023
Arthropathy (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Back disorder (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Back pain (Musculoskeletal and connective tissue disorders) | 12/5013 | 9/5024 | 10/5000 | 15/5023
Bone cyst (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Bone infarction (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Bone pain (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Bursitis (Musculoskeletal and connective tissue disorders) | 0/5013 | 2/5024 | 1/5000 | 1/5023
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/5013 | 2/5024 | 1/5000 | 0/5023
Chondropathy (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 4/5000 | 0/5023
Exostosis (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Fistula (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Fistula discharge (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Flank pain (Musculoskeletal and connective tissue disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Foot deformity (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 3/5000 | 1/5023
Groin pain (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0/5013 | 2/5024 | 1/5000 | 0/5023
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8/5013 | 2/5024 | 10/5000 | 9/5023
Joint effusion (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Knee deformity (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2/5013 | 2/5024 | 3/5000 | 1/5023
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Monarthritis (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3/5013 | 2/5024 | 5/5000 | 4/5023
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3/5013 | 1/5024 | 0/5000 | 2/5023
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 3/5000 | 2/5023
Myalgia (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Myopathy (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Myositis (Musculoskeletal and connective tissue disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Neck mass (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Neck pain (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 2/5000 | 4/5023
Osteitis (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 28/5013 | 23/5024 | 30/5000 | 34/5023
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1/5013 | 1/5024 | 0/5000 | 2/5023
Osteolysis (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0/5013 | 2/5024 | 1/5000 | 2/5023
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7/5013 | 1/5024 | 4/5000 | 2/5023
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Periarthritis (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2/5013 | 1/5024 | 2/5000 | 2/5023
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3/5013 | 3/5024 | 1/5000 | 2/5023
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2/5013 | 3/5024 | 3/5000 | 2/5023
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3/5013 | 2/5024 | 3/5000 | 6/5023
Spondylitis (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Trismus (Musculoskeletal and connective tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Acute megakaryocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Angiosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 1/5024 | 6/5000 | 2/5023
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Benign muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Benign neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/5013 | 5/5024 | 5/5000 | 6/5023
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 4/5023
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 2/5024 | 0/5000 | 3/5023
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 0/5024 | 0/5000 | 1/5023
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/5013 | 5/5024 | 2/5000 | 4/5023
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/5013 | 5/5024 | 9/5000 | 6/5023
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 2/5024 | 2/5000 | 1/5023
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Buccal cavity papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 1/5024 | 0/5000 | 1/5023
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13/5013 | 11/5024 | 4/5000 | 14/5023
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 2/5023
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 2/5023
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/5013 | 4/5024 | 2/5000 | 5/5023
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 2/5024 | 1/5000 | 2/5023
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Genital neoplasm malignant female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 3/5024 | 3/5000 | 0/5023
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 1/5000 | 2/5023
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/5013 | 4/5024 | 3/5000 | 5/5023
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 2/5000 | 0/5023
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 2/5000 | 0/5023
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 3/5024 | 2/5000 | 6/5023
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 3/5000 | 0/5023
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14/5013 | 13/5024 | 21/5000 | 10/5023
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 4/5023
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 2/5024 | 0/5000 | 0/5023
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 2/5023
Malignant neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Malignant nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Maxillofacial sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/5013 | 1/5024 | 4/5000 | 1/5023
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/5013 | 3/5024 | 3/5000 | 1/5023
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/5013 | 5/5024 | 6/5000 | 6/5023
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/5013 | 2/5024 | 2/5000 | 5/5023
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5/5013 | 1/5024 | 2/5000 | 2/5023
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 2/5024 | 0/5000 | 3/5023
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 2/5024 | 1/5000 | 1/5023
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 0/5024 | 1/5000 | 4/5023
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 2/5024 | 0/5000 | 0/5023
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 4/5000 | 4/5023
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 0/5000 | 2/5023
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/5013 | 8/5024 | 2/5000 | 3/5023
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 2/5000 | 0/5023
Peritoneal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Pleura carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12/5013 | 15/5024 | 16/5000 | 12/5023
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 2/5000 | 3/5023
Pseudomyxoma peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 3/5024 | 3/5000 | 4/5023
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 2/5000 | 1/5023
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/5013 | 2/5024 | 0/5000 | 0/5023
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Rhabdomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 2/5023
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 4/5000 | 2/5023
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Tonsillar neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 2/5000 | 0/5023
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Altered state of consciousness (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Amnesia (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Amyotrophic lateral sclerosis (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Anoxic encephalopathy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Aphasia (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Ataxia (Nervous system disorders) | 0/5013 | 2/5024 | 2/5000 | 1/5023
Autonomic nervous system imbalance (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Balance disorder (Nervous system disorders) | 3/5013 | 1/5024 | 1/5000 | 0/5023
Basilar artery stenosis (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Bradykinesia (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Brain mass (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Brain oedema (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Bulbar palsy (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Carotid arteriosclerosis (Nervous system disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Carotid artery aneurysm (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Carotid artery disease (Nervous system disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Carotid artery occlusion (Nervous system disorders) | 1/5013 | 2/5024 | 1/5000 | 0/5023
Carotid artery stenosis (Nervous system disorders) | 26/5013 | 19/5024 | 27/5000 | 20/5023
Carotid artery thrombosis (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Carpal tunnel syndrome (Nervous system disorders) | 1/5013 | 3/5024 | 1/5000 | 3/5023
Central nervous system lesion (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Central pain syndrome (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cerebellar infarction (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Cerebral arteriosclerosis (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cerebral artery embolism (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cerebral artery stenosis (Nervous system disorders) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Cerebral disorder (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Cerebral haemorrhage (Nervous system disorders) | 3/5013 | 0/5024 | 1/5000 | 0/5023
Cerebral infarction (Nervous system disorders) | 1/5013 | 3/5024 | 2/5000 | 2/5023
Cerebral ischaemia (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cerebrovascular accident (Nervous system disorders) | 4/5013 | 7/5024 | 4/5000 | 6/5023
Cerebrovascular disorder (Nervous system disorders) | 0/5013 | 2/5024 | 3/5000 | 2/5023
Cerebrovascular insufficiency (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cervical myelopathy (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Chorea (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Clonic convulsion (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Clonus (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Cognitive disorder (Nervous system disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Coma (Nervous system disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Complex partial seizures (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Consciousness fluctuating (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Convulsion (Nervous system disorders) | 27/5013 | 18/5024 | 23/5000 | 26/5023
Coordination abnormal (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cubital tunnel syndrome (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Dementia (Nervous system disorders) | 2/5013 | 3/5024 | 1/5000 | 3/5023
Dementia Alzheimer's type (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Demyelination (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Depressed level of consciousness (Nervous system disorders) | 0/5013 | 1/5024 | 2/5000 | 1/5023
Diabetic coma (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Diabetic hyperosmolar coma (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 2/5023
Diabetic neuropathy (Nervous system disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Dizziness (Nervous system disorders) | 16/5013 | 19/5024 | 12/5000 | 15/5023
Dizziness postural (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Drug withdrawal convulsions (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Dysarthria (Nervous system disorders) | 2/5013 | 0/5024 | 1/5000 | 3/5023
Dyskinesia (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Dysphasia (Nervous system disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Dysstasia (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Dystonia (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Encephalitis (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Encephalopathy (Nervous system disorders) | 5/5013 | 2/5024 | 2/5000 | 2/5023
Epilepsy (Nervous system disorders) | 18/5013 | 14/5024 | 16/5000 | 7/5023
Facial palsy (Nervous system disorders) | 3/5013 | 4/5024 | 0/5000 | 1/5023
Facial paresis (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Global amnesia (Nervous system disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Grand mal convulsion (Nervous system disorders) | 2/5013 | 4/5024 | 1/5000 | 5/5023
Guillain-Barre syndrome (Nervous system disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Haemorrhage intracranial (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Haemorrhagic transformation stroke (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Head discomfort (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Headache (Nervous system disorders) | 21/5013 | 18/5024 | 16/5000 | 8/5023
Hemiparesis (Nervous system disorders) | 6/5013 | 1/5024 | 1/5000 | 3/5023
Hepatic encephalopathy (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Hyperaesthesia (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Hypersomnia (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hypertensive encephalopathy (Nervous system disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Hypoaesthesia (Nervous system disorders) | 1/5013 | 3/5024 | 4/5000 | 2/5023
Hypoglycaemic coma (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hypoxic encephalopathy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
IIIrd nerve paralysis (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
IVth nerve paralysis (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Intracranial aneurysm (Nervous system disorders) | 0/5013 | 1/5024 | 1/5000 | 2/5023
Intracranial hypotension (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Intracranial pressure increased (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Intraventricular haemorrhage (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Ischaemic neuropathy (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Ischaemic stroke (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lateral medullary syndrome (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lethargy (Nervous system disorders) | 1/5013 | 2/5024 | 0/5000 | 1/5023
Loss of consciousness (Nervous system disorders) | 5/5013 | 1/5024 | 3/5000 | 3/5023
Lumbar radiculopathy (Nervous system disorders) | 2/5013 | 1/5024 | 2/5000 | 0/5023
Memory impairment (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Mental impairment (Nervous system disorders) | 1/5013 | 0/5024 | 2/5000 | 0/5023
Metabolic encephalopathy (Nervous system disorders) | 2/5013 | 0/5024 | 0/5000 | 1/5023
Migraine (Nervous system disorders) | 0/5013 | 2/5024 | 1/5000 | 1/5023
Monoparesis (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Motor neurone disease (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Multiple system atrophy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Muscle spasticity (Nervous system disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Myasthenia gravis (Nervous system disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Myelitis (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Myelopathy (Nervous system disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Myoclonus (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Nerve compression (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Nerve root compression (Nervous system disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Nervous system disorder (Nervous system disorders) | 2/5013 | 0/5024 | 1/5000 | 0/5023
Neuralgia (Nervous system disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Neurological symptom (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Neuromyelitis optica (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Neuropathy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Neuropathy peripheral (Nervous system disorders) | 0/5013 | 2/5024 | 0/5000 | 1/5023
Normal pressure hydrocephalus (Nervous system disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Paraesthesia (Nervous system disorders) | 2/5013 | 2/5024 | 3/5000 | 1/5023
Paraparesis (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Paresis (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Parkinson's disease (Nervous system disorders) | 2/5013 | 1/5024 | 3/5000 | 2/5023
Parkinsonism (Nervous system disorders) | 1/5013 | 2/5024 | 0/5000 | 1/5023
Partial seizures (Nervous system disorders) | 3/5013 | 3/5024 | 0/5000 | 6/5023
Peroneal nerve palsy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pneumocephalus (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Polyneuropathy (Nervous system disorders) | 0/5013 | 0/5024 | 3/5000 | 2/5023
Presyncope (Nervous system disorders) | 2/5013 | 3/5024 | 10/5000 | 4/5023
Radial nerve palsy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Radicular pain (Nervous system disorders) | 0/5013 | 2/5024 | 0/5000 | 1/5023
Radiculitis lumbosacral (Nervous system disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Radiculopathy (Nervous system disorders) | 1/5013 | 0/5024 | 2/5000 | 0/5023
Restless legs syndrome (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Sciatica (Nervous system disorders) | 2/5013 | 1/5024 | 1/5000 | 0/5023
Senile dementia (Nervous system disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Sensory disturbance (Nervous system disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Sensory loss (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Simple partial seizures (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Somnolence (Nervous system disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Speech disorder (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Spinal cord disorder (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Status epilepticus (Nervous system disorders) | 0/5013 | 0/5024 | 1/5000 | 3/5023
Subarachnoid haemorrhage (Nervous system disorders) | 2/5013 | 3/5024 | 3/5000 | 5/5023
Syncope (Nervous system disorders) | 25/5013 | 20/5024 | 31/5000 | 24/5023
Syncope vasovagal (Nervous system disorders) | 3/5013 | 5/5024 | 7/5000 | 3/5023
Temporal lobe epilepsy (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Tension headache (Nervous system disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Tonic convulsion (Nervous system disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Toxic encephalopathy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Transient ischaemic attack (Nervous system disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Tremor (Nervous system disorders) | 1/5013 | 2/5024 | 1/5000 | 0/5023
Trigeminal neuralgia (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Ulnar nerve palsy (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Uraemic encephalopathy (Nervous system disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
VIth nerve paralysis (Nervous system disorders) | 0/5013 | 2/5024 | 0/5000 | 0/5023
Vascular dementia (Nervous system disorders) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Vasculitis cerebral (Nervous system disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Vertebral artery stenosis (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Vertebrobasilar insufficiency (Nervous system disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Wernicke-Korsakoff syndrome (Nervous system disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Abnormal behaviour (Psychiatric disorders) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Acute stress disorder (Psychiatric disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Adjustment disorder (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Adjustment disorder with depressed mood (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Aggression (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Agitation (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Alcohol abuse (Psychiatric disorders) | 3/5013 | 0/5024 | 0/5000 | 1/5023
Alcohol withdrawal syndrome (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Alcoholism (Psychiatric disorders) | 2/5013 | 3/5024 | 0/5000 | 0/5023
Anxiety (Psychiatric disorders) | 4/5013 | 6/5024 | 9/5000 | 2/5023
Anxiety disorder (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Bipolar disorder (Psychiatric disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Completed suicide (Psychiatric disorders) | 1/5013 | 2/5024 | 3/5000 | 2/5023
Confusional state (Psychiatric disorders) | 2/5013 | 6/5024 | 6/5000 | 7/5023
Conversion disorder (Psychiatric disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Delirium (Psychiatric disorders) | 4/5013 | 4/5024 | 1/5000 | 0/5023
Delirium tremens (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Delusion (Psychiatric disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Delusional disorder, persecutory type (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Depressed mood (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Depression (Psychiatric disorders) | 16/5013 | 19/5024 | 11/5000 | 7/5023
Depression suicidal (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Disorientation (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Eating disorder (Psychiatric disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Generalised anxiety disorder (Psychiatric disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hallucination, visual (Psychiatric disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Homicidal ideation (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hypomania (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Impaired self-care (Psychiatric disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Intentional self-injury (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Major depression (Psychiatric disorders) | 2/5013 | 0/5024 | 1/5000 | 0/5023
Mania (Psychiatric disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Mental disorder (Psychiatric disorders) | 0/5013 | 2/5024 | 1/5000 | 1/5023
Mental status changes (Psychiatric disorders) | 9/5013 | 3/5024 | 5/5000 | 4/5023
Nervousness (Psychiatric disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Panic attack (Psychiatric disorders) | 2/5013 | 2/5024 | 0/5000 | 1/5023
Psychiatric symptom (Psychiatric disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Psychotic disorder (Psychiatric disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Sleep disorder (Psychiatric disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Somatisation disorder (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Somatoform disorder (Psychiatric disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Stress (Psychiatric disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Substance abuse (Psychiatric disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Suicidal behaviour (Psychiatric disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Suicidal ideation (Psychiatric disorders) | 3/5013 | 0/5024 | 0/5000 | 0/5023
Suicide attempt (Psychiatric disorders) | 2/5013 | 3/5024 | 1/5000 | 0/5023
Transient psychosis (Psychiatric disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Acute prerenal failure (Renal and urinary disorders) | 1/5013 | 1/5024 | 1/5000 | 1/5023
Anuria (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Azotaemia (Renal and urinary disorders) | 2/5013 | 1/5024 | 0/5000 | 1/5023
Bladder spasm (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Calculus bladder (Renal and urinary disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Calculus ureteric (Renal and urinary disorders) | 1/5013 | 3/5024 | 6/5000 | 1/5023
Calculus urethral (Renal and urinary disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Calculus urinary (Renal and urinary disorders) | 0/5013 | 2/5024 | 2/5000 | 2/5023
Cystitis haemorrhagic (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Diabetic cystopathy (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Diabetic nephropathy (Renal and urinary disorders) | 1/5013 | 1/5024 | 0/5000 | 2/5023
Dysuria (Renal and urinary disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Glomerulonephritis chronic (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Haematuria (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hydronephrosis (Renal and urinary disorders) | 3/5013 | 4/5024 | 3/5000 | 0/5023
Hydroureter (Renal and urinary disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Incontinence (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Kidney enlargement (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Micturition disorder (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Nephritis autoimmune (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Nephritis interstitial (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Nephrolithiasis (Renal and urinary disorders) | 4/5013 | 9/5024 | 5/5000 | 4/5023
Nephropathy (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Nephropathy toxic (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Nephrotic syndrome (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Neurogenic bladder (Renal and urinary disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Obstructive uropathy (Renal and urinary disorders) | 0/5013 | 2/5024 | 0/5000 | 0/5023
Perinephric effusion (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Pollakiuria (Renal and urinary disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Proteinuria (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 2/5023
Pyelectasia (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pyuria (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Renal artery stenosis (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Renal colic (Renal and urinary disorders) | 1/5013 | 3/5024 | 2/5000 | 1/5023
Renal cyst (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Renal embolism (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Renal failure (Renal and urinary disorders) | 8/5013 | 9/5024 | 11/5000 | 7/5023
Renal failure acute (Renal and urinary disorders) | 33/5013 | 24/5024 | 32/5000 | 12/5023
Renal failure chronic (Renal and urinary disorders) | 2/5013 | 6/5024 | 4/5000 | 2/5023
Renal impairment (Renal and urinary disorders) | 2/5013 | 3/5024 | 4/5000 | 3/5023
Renal mass (Renal and urinary disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Residual urine (Renal and urinary disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Single functional kidney (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Stress urinary incontinence (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Tubulointerstitial nephritis (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Ureteric obstruction (Renal and urinary disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Ureteric stenosis (Renal and urinary disorders) | 2/5013 | 0/5024 | 1/5000 | 0/5023
Urethral disorder (Renal and urinary disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Urethral meatus stenosis (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Urethral polyp (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Urethral stenosis (Renal and urinary disorders) | 1/5013 | 1/5024 | 0/5000 | 2/5023
Urinary bladder polyp (Renal and urinary disorders) | 2/5013 | 0/5024 | 0/5000 | 2/5023
Urinary incontinence (Renal and urinary disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Urinary retention (Renal and urinary disorders) | 6/5013 | 4/5024 | 8/5000 | 4/5023
Urinary tract disorder (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Urinary tract obstruction (Renal and urinary disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Urine flow decreased (Renal and urinary disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Balanitis (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Bartholin's cyst (Reproductive system and breast disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 9/5013 | 9/5024 | 17/5000 | 13/5023
Breast mass (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Breast microcalcification (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cervical dysplasia (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cystocele (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Epididymitis (Reproductive system and breast disorders) | 2/5013 | 2/5024 | 0/5000 | 1/5023
Genital prolapse (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Genital ulceration (Reproductive system and breast disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Ovarian cyst (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Pelvic pain (Reproductive system and breast disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Prostatic obstruction (Reproductive system and breast disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Prostatism (Reproductive system and breast disorders) | 2/5013 | 1/5024 | 1/5000 | 0/5023
Prostatitis (Reproductive system and breast disorders) | 1/5013 | 3/5024 | 0/5000 | 3/5023
Prostatomegaly (Reproductive system and breast disorders) | 1/5013 | 4/5024 | 2/5000 | 0/5023
Rectocele (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Uterine cyst (Reproductive system and breast disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Uterine prolapse (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 1/5000 | 2/5023
Uterovaginal prolapse (Reproductive system and breast disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Vaginal prolapse (Reproductive system and breast disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Varicocele (Reproductive system and breast disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 2/5000 | 2/5023
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3/5013 | 0/5024 | 1/5000 | 1/5023
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 1/5024 | 1/5000 | 2/5023
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 3/5013 | 1/5024 | 1/5000 | 1/5023
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 2/5000 | 0/5023
Asthma (Respiratory, thoracic and mediastinal disorders) | 2/5013 | 2/5024 | 2/5000 | 5/5023
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2/5013 | 0/5024 | 0/5000 | 0/5023
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 1/5024 | 1/5000 | 2/5023
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Choking (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 2/5000 | 1/5023
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14/5013 | 13/5024 | 21/5000 | 17/5023
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cough (Respiratory, thoracic and mediastinal disorders) | 2/5013 | 0/5024 | 0/5000 | 3/5023
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14/5013 | 8/5024 | 14/5000 | 13/5023
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2/5013 | 1/5024 | 2/5000 | 2/5023
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 2/5024 | 0/5000 | 0/5023
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 1/5024 | 0/5000 | 1/5023
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 1/5000 | 1/5023
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5/5013 | 5/5024 | 5/5000 | 5/5023
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2/5013 | 1/5024 | 1/5000 | 0/5023
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 2/5024 | 0/5000 | 0/5023
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 12/5013 | 10/5024 | 7/5000 | 5/5023
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2/5013 | 4/5024 | 0/5000 | 0/5023
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 2/5024 | 0/5000 | 1/5023
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 2/5024 | 1/5000 | 1/5023
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1/5013 | 1/5024 | 2/5000 | 1/5023
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8/5013 | 7/5024 | 10/5000 | 9/5023
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4/5013 | 0/5024 | 2/5000 | 4/5023
Angioedema (Skin and subcutaneous tissue disorders) | 1/5013 | 1/5024 | 3/5000 | 1/5023
Blister (Skin and subcutaneous tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1/5013 | 1/5024 | 3/5000 | 0/5023
Dermal cyst (Skin and subcutaneous tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Ecchymosis (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Eczema (Skin and subcutaneous tissue disorders) | 1/5013 | 0/5024 | 2/5000 | 1/5023
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Night sweats (Skin and subcutaneous tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Pruritus (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Psoriasis (Skin and subcutaneous tissue disorders) | 1/5013 | 0/5024 | 0/5000 | 1/5023
Purpura (Skin and subcutaneous tissue disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Rash (Skin and subcutaneous tissue disorders) | 1/5013 | 3/5024 | 0/5000 | 0/5023
Rash erythematous (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Scar (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 3/5023
Segmented hyalinising vasculitis (Skin and subcutaneous tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Skin discolouration (Skin and subcutaneous tissue disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Skin oedema (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Skin ulcer (Skin and subcutaneous tissue disorders) | 3/5013 | 5/5024 | 1/5000 | 5/5023
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Urticaria (Skin and subcutaneous tissue disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Cardiac assistance device user (Social circumstances) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Elderly (Social circumstances) | 1/5013 | 1/5024 | 0/5000 | 0/5023
Social problem (Social circumstances) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Social stay hospitalisation (Social circumstances) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Alcohol detoxification (Surgical and medical procedures) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Angioplasty (Surgical and medical procedures) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Bile duct stent insertion (Surgical and medical procedures) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Blepharoplasty (Surgical and medical procedures) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Carotid endarterectomy (Surgical and medical procedures) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Cataract operation (Surgical and medical procedures) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Cholecystectomy (Surgical and medical procedures) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Coronary angioplasty (Surgical and medical procedures) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Finger amputation (Surgical and medical procedures) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Plasmapheresis (Surgical and medical procedures) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Removal of internal fixation (Surgical and medical procedures) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Splenectomy (Surgical and medical procedures) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Accelerated hypertension (Vascular disorders) | 1/5013 | 3/5024 | 2/5000 | 1/5023
Aneurysm (Vascular disorders) | 1/5013 | 1/5024 | 1/5000 | 0/5023
Angiopathy (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Aortic aneurysm (Vascular disorders) | 5/5013 | 8/5024 | 8/5000 | 4/5023
Aortic aneurysm rupture (Vascular disorders) | 0/5013 | 0/5024 | 2/5000 | 2/5023
Aortic arteriosclerosis (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Aortic dissection (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Aortic embolus (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Aortic rupture (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Aortic stenosis (Vascular disorders) | 1/5013 | 1/5024 | 0/5000 | 3/5023
Arterial occlusive disease (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Arterial restenosis (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Arterial rupture (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Arterial stenosis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Arteriosclerosis (Vascular disorders) | 2/5013 | 3/5024 | 4/5000 | 3/5023
Arteriosclerosis obliterans (Vascular disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Arteritis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Blood pressure inadequately controlled (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 1/5023
Cardiovascular insufficiency (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Circulatory collapse (Vascular disorders) | 2/5013 | 0/5024 | 1/5000 | 1/5023
Deep vein thrombosis (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Diabetic macroangiopathy (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Diabetic vascular disorder (Vascular disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Embolism (Vascular disorders) | 1/5013 | 0/5024 | 0/5000 | 0/5023
Essential hypertension (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 2/5023
Extremity necrosis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Femoral arterial stenosis (Vascular disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Femoral artery occlusion (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Fibromuscular dysplasia (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Haematoma (Vascular disorders) | 2/5013 | 1/5024 | 1/5000 | 1/5023
Haemorrhage (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Hypertension (Vascular disorders) | 14/5013 | 15/5024 | 19/5000 | 20/5023
Hypertensive crisis (Vascular disorders) | 7/5013 | 3/5024 | 7/5000 | 12/5023
Hypertensive emergency (Vascular disorders) | 2/5013 | 0/5024 | 1/5000 | 0/5023
Hypotension (Vascular disorders) | 19/5013 | 8/5024 | 26/5000 | 9/5023
Hypovolaemic shock (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Iliac artery stenosis (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Intermittent claudication (Vascular disorders) | 2/5013 | 1/5024 | 0/5000 | 0/5023
Ischaemia (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Lymphoedema (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Malignant hypertension (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Orthostatic hypotension (Vascular disorders) | 3/5013 | 6/5024 | 7/5000 | 7/5023
Peripheral arterial occlusive disease (Vascular disorders) | 0/5013 | 1/5024 | 1/5000 | 1/5023
Peripheral artery aneurysm (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Peripheral ischaemia (Vascular disorders) | 1/5013 | 0/5024 | 1/5000 | 0/5023
Peripheral vascular disorder (Vascular disorders) | 1/5013 | 5/5024 | 0/5000 | 1/5023
Phlebitis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Post thrombotic syndrome (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Shock (Vascular disorders) | 0/5013 | 1/5024 | 1/5000 | 0/5023
Subclavian artery stenosis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 1/5023
Superior vena caval occlusion (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
Temporal arteritis (Vascular disorders) | 1/5013 | 4/5024 | 0/5000 | 0/5023
Thrombophlebitis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Thrombophlebitis superficial (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Thrombosis (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Varicose vein (Vascular disorders) | 0/5013 | 1/5024 | 1/5000 | 2/5023
Vascular pseudoaneurysm (Vascular disorders) | 1/5013 | 0/5024 | 2/5000 | 0/5023
Vasculitis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Venous stasis (Vascular disorders) | 0/5013 | 0/5024 | 0/5000 | 1/5023
Venous thrombosis (Vascular disorders) | 0/5013 | 0/5024 | 1/5000 | 0/5023
Venous thrombosis limb (Vascular disorders) | 0/5013 | 1/5024 | 0/5000 | 0/5023
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Aspirin + Extended Release Dipyridamole / Telmisartan | Aspirin + Extended Release Dipyridamole / Placebo | Clopidogrel / Telmisartan | Clopidogrel / Placebo
Headache (leading to permanent discont. of study medication) (Nervous system disorders) | 318/5013 | 280/5024 | 42/5000 | 50/5023
Dizziness or lightheadedness (Solicited question at Day 7) (Nervous system disorders) | 768/5086 | 597/5095 | 510/5060 | 398/5091
Headache (Solicited question at Day 7) (Nervous system disorders) | 1515/5086 | 1556/5095 | 491/5060 | 546/5091

LIMITATIONS AND CAVEATS:
All SAEs and AEs that led to temporary or permanent trial drug discontinuation were reported, except in Japan, where all AEs were collected. Protocol-defined outcome events were not reported as AEs, but were recorded on the appropriate form

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.